CLINICAL TRIAL: NCT00137111
Title: Total XV - Total Therapy Study XV for Newly Diagnosed Patients With Acute Lymphoblastic Leukemia
Brief Title: Therapy for Newly Diagnosed Patients With Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TOTXV; R37CA036401 (NIH); P30CA021765 (NIH); F32CA141762 (NIH)
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Results first posted 2011-04-26 (Estimated); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Lymphoblastic Leukemia, Acute
Keywords: Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia | interventions — Prednisone; Dexamethasone; Vincristine; Daunorubicin; Doxorubicin; Asparaginase; pegaspargase; asparaginase erwinia chrysanthemi recombinant; Methotrexate; Cyclophosphamide; Cytarabine; Etoposide; Mercaptopurine; Imatinib Mesylate; Drug Therapy; Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1 (Other)
  Interventions: Drug: Prednisone, Dexamethasone, Vincristine, Daunorubicin; Drug: Doxorubicin, L-asparaginase, PEG-L-asparaginase, Erwinia asparaginase; Drug: Methotrexate, Cyclophosphamide, Cytarabine, Etoposide; Drug: Mercaptopurine, Imatinib; Procedure: chemotherapy, intrathecal chemotherapy; Procedure: steroid therapy, hematopoietic stem cell transplantation
- 2 (Other)
  Interventions: Drug: Prednisone, Dexamethasone, Vincristine, Daunorubicin; Drug: Doxorubicin, L-asparaginase, PEG-L-asparaginase, Erwinia asparaginase; Drug: Methotrexate, Cyclophosphamide, Cytarabine, Etoposide; Drug: Mercaptopurine, Imatinib; Procedure: chemotherapy, intrathecal chemotherapy; Procedure: steroid therapy, hematopoietic stem cell transplantation

INTERVENTIONS:
Drug: Prednisone, Dexamethasone, Vincristine, Daunorubicin — See Detailed Description sections for details on treatment interventions.
Drug: Doxorubicin, L-asparaginase, PEG-L-asparaginase, Erwinia asparaginase — See Detailed Description sections for details on treatment interventions.
Drug: Methotrexate, Cyclophosphamide, Cytarabine, Etoposide — See Detailed Description sections for details on treatment interventions.
Drug: Mercaptopurine, Imatinib — See Detailed Description sections for details on treatment interventions.
Procedure: chemotherapy, intrathecal chemotherapy — See Detailed Description sections for details on treatment interventions.
Procedure: steroid therapy, hematopoietic stem cell transplantation — See Detailed Description sections for details on treatment interventions.

SUMMARY:
The primary objective is to estimate the overall event-free survival of children at least one year of age at diagnosis who are treated with risk-directed therapy and to monitor the molecular remission induction rate.

DETAILED DESCRIPTION:
These are the following secondary objectives:

* To determine if CNS irradiation can be safely omitted in the context of the systemic therapy used in the protocol.
* To identify whether prolonged (24 hour) intravenous infusions of HDMTX produce greater methotrexate polyglutamate (MTXPG) accumulation than short (4 hour) infusions 42 hours after 1 gm/m2 of HDMTX, stratified for lineage (T- vs B-lineage) and ploidy (hyperdiploid vs non-hyperdiploid B-lineage).
* To determine whether prolonged (24 hour) intravenous infusions of HDMTX produce greater antileukemic effects than short (4 hour) infusions, based on the inhibition of de novo purine synthesis in bone marrow blasts and the decrease in circulating blasts during the 4 day "window" prior to initiation of conventional remission induction therapy.
* MRD
* Other exploratory objectives

Details of Treatment Plan

Treatment will consist of three main phases, Remission Induction, Consolidation, and Continuation. Treatment with an Upfront HDMTX Window for research purposes will be optional.

All patients will receive IT therapy on day 1, dose is age dependent.

Upfront High-Dose Methotrexate Window

HDMTX (1 g/m2) as a 4 hour infusion versus as a 24 hour infusion. Leucovorin rescue will be given.

Remission Induction

Prednisone 40 mg/m2/day PO Days 5 - 32 Vincristine 1.5 mg/m2/week IV Days 5, 12, 19, 26 Daunorubicin 25 mg/m2/week IV Days 5, 12 L-asparaginase 10,000 Unit/m2/dose IM Days 6, 8, 10, 12, 14, 16 (19, 21, 23) Cyclophosphamide 1000 mg/m2/dose IV Day 26 Cytarabine 75 mg/m2/dose IV Days 27-30, 34-37 6-Mercaptopurine 60 mg/m2/dose PO Days 26-39 Imatinib 40 mg/m2 bid for Ph positive patients starting Day 22 of induction. Intrathecal therapy will be administered on day 1 and 19, dose age dependent. Patients with high risk of CNS relapse will receive additional IT treatments on days 8 and 26.

Consolidation Treatment

High dose methotrexate targeted dose depending on risk status, days 1, 15, 29, and 43 and mercaptopurine 50 mg/m2/day, days 1-56.

Reintensification treatment for patients with high risk disease:

Patients with high risk disease will be offered the option of hematopoietic stem cell transplant (HSCT) and may receive an additional 1-2 cycles of reintensification treatment prior to maximize the anti-leukemic kill before transplant.

Dexamethasone 20 mg/m2 PO days 1-3 Cytarabine 2 g/m2 IV x 4 doses, days 3-5 Etoposide 100 mg/m2 IV x 5 doses, days 3-5 L-asparaginase 25,000 Units/m2 IM day 6 Intrathecal treatment Day 5

Continuation Treatment (lasts 120 weeks for girls and 146 weeks for boys)

Treatment will depend on risk classification: low versus standard versus high risk

Treatment weeks 1 to 20:

Week Standard/High Risk Low Risk

1. DEX + DOX + VCR + 6MP + ASP 6MP + DEX + VCR
2. 6MP + ASP 6MP + MTX
3. 6MP + ASP 6MP + MTX
4. DEX + DOX + VCR + 6MP + ASP 6MP + DEX + VCR
5. 6MP + ASP 6MP + MTX
6. 6MP + ASP 6MP + MTX
7. Reinduction I§ Reinduction I
8. Reinduction I Reinduction I
9. Reinduction I Reinduction I
10. 6MP + ASP 6MP + MTX
11. DOX + VCR + 6MP + ASP 6MP + MTX
12. 6MP + ASP 6MP + MTX
13. 6MP + ASP 6MP + MTX
14. DEX + DOX + VCR + 6MP + ASP 6MP + DEX + VCR
15. 6MP + ASP 6MP + MTX
16. 6MP + ASP 6MP + MTX
17. Reinduction II Reinduction II
18. Reinduction II Reinduction II
19. Reinduction II Reinduction II
20. No chemotherapy 6MP + MTX

    Dexamethasone 12 mg/m2 (std/high risk) or 8 mg/m2 (low risk) PO daily (tid) x 5 days, Days 1-5 Doxorubicin 30 mg/m2 IV, Day 1 Vincristine 2.0 mg/m2 IV push (max. 2 mg), Day 1 Mercaptopurine 50 mg/m2 PO daily x 7 days (std/high risk), Days 1-7 75 mg/m2 PO daily x 7 days (low risk), Days 1-7 L-asparaginase 25,000 Unit/m2 IM, Day 1 Methotrexate 40 mg/m2 IV or IM, Day 1

    Reinduction I and II

    This phase of treatment will be started at weeks 7 and 17 after bone marrow examination confirms complete remission. Reinduction treatment will be given twice: weeks 7 to 9 and weeks 17 to 19 for all patients.

    Reinduction I for Standard/High Risk ALL:

    Dexamethasone 8 mg/m2/day PO (t.i.d.) Days 1-8, 15, 21, Vincristine 1.5 mg/m2/week IV (max 2 mg) Days 1, 8, 15, Doxorubicin 30 mg/m2 Days 1, 8, L-asparaginase 25,000 Unit/m2 IM Days 1, 8, 15, Intrathecal chemotherapy, dose age dependent Day 1.

    Reinduction II for Standard/High Risk ALL:

    Dexamethasone 8 mg/m2/day PO (t.i.d.) Days 1-8, 15-21, Vincristine 1.5 mg/m2/week IV (max 2 mg) Days 1, 8, 15, L-asparaginase 25,000 Unit/m2, weekly IM Days 1, 8, 17, Intrathecal chemotherapy, dose age dependent Day 1 High-dose cytarabine 2 gm/m2 IV q 12 Days 15, 16

    Reinduction I and II for Low Risk ALL Dexamethasone 8 mg/m2/day PO (t.i.d.) Days 1-8, 15-21 Vincristine 1.5 mg/m2/week IV (max 2 mg), Days 1, 8, 15 L-asparaginase 10,000 Unit/m2/thrice weekly IM Days 2, 4, 6, 8, 10, 12, 15, 17, 19 Doxorubicin 30 mg/m2/week IV Day 1 Intrathecal chemotherapy, dose age dependent on Day 1

    Treatment Weeks 21 to end of therapy Week Standard/High Risk Low Risk
21. 6MP + MTX 6MP + MTX
22. 6MP + MTX 6MP + MTX
23. Cyclo + Ara-C 6MP + MTX
24. DEX + VCR 6MP + DEX + VCR
25. 6MP + MTX 6MP + MTX
26. 6MP + MTX 6MP + MTX
27. Cyclo + Ara-C 6MP + MTX
28. DEX + VCR 6MP + DEX + VCR

Mercaptopurine 75 mg/m2 PO, daily x 7 days, Days 1-7 Methotrexate 40 mg/m2 IV or IM, Day 1 Cyclophosphamide 300 mg/m2 IV, Day 1 Cytarabine 300 mg/m2 IV, Day 1 Dexamethasone 12 mg/m2 (std/high risk) or 8 mg/m2 (low risk) PO daily (tid) x 5, Day 1-5 Vincristine 2.0 mg/m2 IV push (max. 2 mg), Day 1

The same treatment (weeks 21-28) will be repeated for a total of 6 times (until week 68). After week 68, all patients will receive daily 6MP and weekly MTX with pulses of dexamethasone and vincristine every 4 weeks until week 100, after which only 6MP and methotrexate will be given. Intrathecal treatment will be given every 8 weeks only to patients at high risk of CNS relapse after week 48 and will be discontinued after week 96. Continuation therapy will be discontinued after 120 weeks in girls and after 146 weeks in boys

Patients who meet the criteria of high-risk ALL are candidates for allogeneic hematopoietic stem cell transplantation. However, if the option is declined by the patients or guardians, or the procedure is deemed unsuitable by the attending physician and the principal investigator, the patient will remain on study and continue to receive chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-B-cell ALL by immunophenotyping, as determined by the reactivity pattern to a panel of monoclonal antibodies with flow cytometry as well as morphology and cytochemical staining.
* Age range: 1 to 18 years (inclusive).

Exclusion Criteria:

• Previously treated with chemotherapy for one week or longer.

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 501 (Actual)
Dates: Start 2000-07-08 (Actual); Primary Completion 2010-11 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Hon Pui, M.D., Principal Investigator — St. Jude Children's Research Hospital
Locations (2):
- United States (2):
  - St Jude Children's Research Hospital, Memphis, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas

REFERENCES:
- [Background] Yeoh EJ, Ross ME, Shurtleff SA, Williams WK, Patel D, Mahfouz R, Behm FG, Raimondi SC, Relling MV, Patel A, Cheng C, Campana D, Wilkins D, Zhou X, Li J, Liu H, Pui CH, Evans WE, Naeve C, Wong L, Downing JR. Classification, subtype discovery, and prediction of outcome in pediatric acute lymphoblastic leukemia by gene expression profiling. Cancer Cell. 2002 Mar;1(2):133-43. doi: 10.1016/s1535-6108(02)00032-6. PMID 12086872
- [Background] Coustan-Smith E, Sancho J, Hancock ML, Razzouk BI, Ribeiro RC, Rivera GK, Rubnitz JE, Sandlund JT, Pui CH, Campana D. Use of peripheral blood instead of bone marrow to monitor residual disease in children with acute lymphoblastic leukemia. Blood. 2002 Oct 1;100(7):2399-402. doi: 10.1182/blood-2002-04-1130. PMID 12239148
- [Background] Cheok MH, Yang W, Pui CH, Downing JR, Cheng C, Naeve CW, Relling MV, Evans WE. Treatment-specific changes in gene expression discriminate in vivo drug response in human leukemia cells. Nat Genet. 2003 May;34(1):85-90. doi: 10.1038/ng1151. PMID 12704389
- [Background] Neale GA, Coustan-Smith E, Stow P, Pan Q, Chen X, Pui CH, Campana D. Comparative analysis of flow cytometry and polymerase chain reaction for the detection of minimal residual disease in childhood acute lymphoblastic leukemia. Leukemia. 2004 May;18(5):934-8. doi: 10.1038/sj.leu.2403348. PMID 15029212
- [Background] Pauley JL, Panetta JC, Schmidt J, Kornegay N, Relling MV, Pui CH. Late-onset delayed excretion of methotrexate. Cancer Chemother Pharmacol. 2004 Aug;54(2):146-52. doi: 10.1007/s00280-004-0797-y. Epub 2004 May 18. PMID 15148625
- [Background] Pui CH, Relling MV, Sandlund JT, Downing JR, Campana D, Evans WE. Rationale and design of Total Therapy Study XV for newly diagnosed childhood acute lymphoblastic leukemia. Ann Hematol. 2004;83 Suppl 1:S124-6. doi: 10.1007/s00277-004-0850-2. PMID 15124703
- [Background] Cheng Q, Wu B, Kager L, Panetta JC, Zheng J, Pui CH, Relling MV, Evans WE. A substrate specific functional polymorphism of human gamma-glutamyl hydrolase alters catalytic activity and methotrexate polyglutamate accumulation in acute lymphoblastic leukaemia cells. Pharmacogenetics. 2004 Aug;14(8):557-67. doi: 10.1097/01.fpc.0000114761.78957.7e. PMID 15284538
- [Background] Zaza G, Yang W, Kager L, Cheok M, Downing J, Pui CH, Cheng C, Relling MV, Evans WE. Acute lymphoblastic leukemia with TEL-AML1 fusion has lower expression of genes involved in purine metabolism and lower de novo purine synthesis. Blood. 2004 Sep 1;104(5):1435-41. doi: 10.1182/blood-2003-12-4306. Epub 2004 May 13. PMID 15142881
- [Background] Hijiya N, Onciu M, Howard SC, Zhang Z, Cheng C, Sandlund JT, Kyzer EP, Behm FG, Pui CH. Utility of automated counting to determine absolute neutrophil counts and absolute phagocyte counts for pediatric cancer treatment protocols. Cancer. 2004 Dec 1;101(11):2681-6. doi: 10.1002/cncr.20677. PMID 15517573
- [Background] Kager L, Cheok M, Yang W, Zaza G, Cheng Q, Panetta JC, Pui CH, Downing JR, Relling MV, Evans WE. Folate pathway gene expression differs in subtypes of acute lymphoblastic leukemia and influences methotrexate pharmacodynamics. J Clin Invest. 2005 Jan;115(1):110-7. doi: 10.1172/JCI22477. PMID 15630450
- [Background] Lowe EJ, Pui CH, Hancock ML, Geiger TL, Khan RB, Sandlund JT. Early complications in children with acute lymphoblastic leukemia presenting with hyperleukocytosis. Pediatr Blood Cancer. 2005 Jul;45(1):10-5. doi: 10.1002/pbc.20178. PMID 15547931
- [Background] McCarville MB, Adelman CS, Li C, Xiong X, Furman WL, Razzouk BI, Pui CH, Sandlund JT. Typhlitis in childhood cancer. Cancer. 2005 Jul 15;104(2):380-7. doi: 10.1002/cncr.21134. PMID 15952190
- [Background] Cheng Q, Yang W, Raimondi SC, Pui CH, Relling MV, Evans WE. Karyotypic abnormalities create discordance of germline genotype and cancer cell phenotypes. Nat Genet. 2005 Aug;37(8):878-82. doi: 10.1038/ng1612. Epub 2005 Jul 24. PMID 16041371
- [Background] Pui CH, Evans WE. Treatment of acute lymphoblastic leukemia. N Engl J Med. 2006 Jan 12;354(2):166-78. doi: 10.1056/NEJMra052603. No abstract available. PMID 16407512
- [Background] Coustan-Smith E, Ribeiro RC, Stow P, Zhou Y, Pui CH, Rivera GK, Pedrosa F, Campana D. A simplified flow cytometric assay identifies children with acute lymphoblastic leukemia who have a superior clinical outcome. Blood. 2006 Jul 1;108(1):97-102. doi: 10.1182/blood-2006-01-0066. Epub 2006 Mar 14. PMID 16537802
- [Background] Flotho C, Coustan-Smith E, Pei D, Iwamoto S, Song G, Cheng C, Pui CH, Downing JR, Campana D. Genes contributing to minimal residual disease in childhood acute lymphoblastic leukemia: prognostic significance of CASP8AP2. Blood. 2006 Aug 1;108(3):1050-7. doi: 10.1182/blood-2006-01-0322. Epub 2006 Apr 20. PMID 16627760
- [Background] Karimova EJ, Rai SN, Ingle D, Ralph AC, Deng X, Neel MD, Howard SC, Pui CH, Kaste SC. MRI of knee osteonecrosis in children with leukemia and lymphoma: Part 2, clinical and imaging patterns. AJR Am J Roentgenol. 2006 Feb;186(2):477-82. doi: 10.2214/AJR.04.1597. PMID 16423956
- [Background] Cheng Q, Cheng C, Crews KR, Ribeiro RC, Pui CH, Relling MV, Evans WE. Epigenetic regulation of human gamma-glutamyl hydrolase activity in acute lymphoblastic leukemia cells. Am J Hum Genet. 2006 Aug;79(2):264-74. doi: 10.1086/505645. Epub 2006 Jun 6. PMID 16826517
- [Background] Mullighan CG, Goorha S, Radtke I, Miller CB, Coustan-Smith E, Dalton JD, Girtman K, Mathew S, Ma J, Pounds SB, Su X, Pui CH, Relling MV, Evans WE, Shurtleff SA, Downing JR. Genome-wide analysis of genetic alterations in acute lymphoblastic leukaemia. Nature. 2007 Apr 12;446(7137):758-64. doi: 10.1038/nature05690. PMID 17344859
- [Background] Hinds PS, Burghen EA, Zhou Y, Zhang L, West N, Bashore L, Pui CH. The Health Utilities Index 3 invalidated when completed by nurses for pediatric oncology patients. Cancer Nurs. 2007 May-Jun;30(3):169-77. doi: 10.1097/01.NCC.0000270700.11425.4d. PMID 17510579
- [Background] Karimova EJ, Rai SN, Howard SC, Neel M, Britton L, Pui CH, Kaste SC. Femoral head osteonecrosis in pediatric and young adult patients with leukemia or lymphoma. J Clin Oncol. 2007 Apr 20;25(12):1525-31. doi: 10.1200/JCO.2006.07.9947. PMID 17442995
- [Background] Flotho C, Coustan-Smith E, Pei D, Cheng C, Song G, Pui CH, Downing JR, Campana D. A set of genes that regulate cell proliferation predicts treatment outcome in childhood acute lymphoblastic leukemia. Blood. 2007 Aug 15;110(4):1271-7. doi: 10.1182/blood-2007-01-068478. Epub 2007 Apr 24. PMID 17456722
- [Background] Hinds PS, Hockenberry MJ, Gattuso JS, Srivastava DK, Tong X, Jones H, West N, McCarthy KS, Sadeh A, Ash M, Fernandez C, Pui CH. Dexamethasone alters sleep and fatigue in pediatric patients with acute lymphoblastic leukemia. Cancer. 2007 Nov 15;110(10):2321-30. doi: 10.1002/cncr.23039. PMID 17926333
- [Background] Marchese VG, Connolly BH, Able C, Booten AR, Bowen P, Porter BM, Rai SN, Hancock ML, Pui CH, Howard S, Neel MD, Kaste SC. Relationships among severity of osteonecrosis, pain, range of motion, and functional mobility in children, adolescents, and young adults with acute lymphoblastic leukemia. Phys Ther. 2008 Mar;88(3):341-50. doi: 10.2522/ptj.20070108. Epub 2008 Jan 17. PMID 18202079
- [Background] Pui CH, Robison LL, Look AT. Acute lymphoblastic leukaemia. Lancet. 2008 Mar 22;371(9617):1030-43. doi: 10.1016/S0140-6736(08)60457-2. PMID 18358930
- [Background] Sorich MJ, Pottier N, Pei D, Yang W, Kager L, Stocco G, Cheng C, Panetta JC, Pui CH, Relling MV, Cheok MH, Evans WE. In vivo response to methotrexate forecasts outcome of acute lymphoblastic leukemia and has a distinct gene expression profile. PLoS Med. 2008 Apr 15;5(4):e83. doi: 10.1371/journal.pmed.0050083. PMID 18416598
- [Background] Yang L, Panetta JC, Cai X, Yang W, Pei D, Cheng C, Kornegay N, Pui CH, Relling MV. Asparaginase may influence dexamethasone pharmacokinetics in acute lymphoblastic leukemia. J Clin Oncol. 2008 Apr 20;26(12):1932-9. doi: 10.1200/JCO.2007.13.8404. PMID 18421047
- [Background] Mullighan CG, Miller CB, Radtke I, Phillips LA, Dalton J, Ma J, White D, Hughes TP, Le Beau MM, Pui CH, Relling MV, Shurtleff SA, Downing JR. BCR-ABL1 lymphoblastic leukaemia is characterized by the deletion of Ikaros. Nature. 2008 May 1;453(7191):110-4. doi: 10.1038/nature06866. Epub 2008 Apr 13. PMID 18408710
- [Background] French D, Yang W, Hamilton LH, Neale G, Fan Y, Downing JR, Cox NJ, Pui CH, Evans WE, Relling MV. Concordant gene expression in leukemia cells and normal leukocytes is associated with germline cis-SNPs. PLoS One. 2008 May 14;3(5):e2144. doi: 10.1371/journal.pone.0002144. PMID 18478092
- [Background] Kamdem LK, Hamilton L, Cheng C, Liu W, Yang W, Johnson JA, Pui CH, Relling MV. Genetic predictors of glucocorticoid-induced hypertension in children with acute lymphoblastic leukemia. Pharmacogenet Genomics. 2008 Jun;18(6):507-14. doi: 10.1097/FPC.0b013e3282fc5801. PMID 18496130
- [Background] Yang JJ, Bhojwani D, Yang W, Cai X, Stocco G, Crews K, Wang J, Morrison D, Devidas M, Hunger SP, Willman CL, Raetz EA, Pui CH, Evans WE, Relling MV, Carroll WL. Genome-wide copy number profiling reveals molecular evolution from diagnosis to relapse in childhood acute lymphoblastic leukemia. Blood. 2008 Nov 15;112(10):4178-83. doi: 10.1182/blood-2008-06-165027. Epub 2008 Sep 2. PMID 18768390
- [Background] Roberson JR, Raju S, Shelso J, Pui CH, Howard SC. Diabetic ketoacidosis during therapy for pediatric acute lymphoblastic leukemia. Pediatr Blood Cancer. 2008 Jun;50(6):1207-12. doi: 10.1002/pbc.21505. PMID 18266226
- [Background] Mullighan CG, Su X, Zhang J, Radtke I, Phillips LA, Miller CB, Ma J, Liu W, Cheng C, Schulman BA, Harvey RC, Chen IM, Clifford RJ, Carroll WL, Reaman G, Bowman WP, Devidas M, Gerhard DS, Yang W, Relling MV, Shurtleff SA, Campana D, Borowitz MJ, Pui CH, Smith M, Hunger SP, Willman CL, Downing JR; Children's Oncology Group. Deletion of IKZF1 and prognosis in acute lymphoblastic leukemia. N Engl J Med. 2009 Jan 29;360(5):470-80. doi: 10.1056/NEJMoa0808253. Epub 2009 Jan 7. PMID 19129520
- [Background] Yang JJ, Cheng C, Yang W, Pei D, Cao X, Fan Y, Pounds SB, Neale G, Trevino LR, French D, Campana D, Downing JR, Evans WE, Pui CH, Devidas M, Bowman WP, Camitta BM, Willman CL, Davies SM, Borowitz MJ, Carroll WL, Hunger SP, Relling MV. Genome-wide interrogation of germline genetic variation associated with treatment response in childhood acute lymphoblastic leukemia. JAMA. 2009 Jan 28;301(4):393-403. doi: 10.1001/jama.2009.7. PMID 19176441
- [Background] Coustan-Smith E, Mullighan CG, Onciu M, Behm FG, Raimondi SC, Pei D, Cheng C, Su X, Rubnitz JE, Basso G, Biondi A, Pui CH, Downing JR, Campana D. Early T-cell precursor leukaemia: a subtype of very high-risk acute lymphoblastic leukaemia. Lancet Oncol. 2009 Feb;10(2):147-56. doi: 10.1016/S1470-2045(08)70314-0. Epub 2009 Jan 13. PMID 19147408
- [Background] Roberson JR, Spraker HL, Shelso J, Zhou Y, Inaba H, Metzger ML, Rubnitz JE, Ribeiro RC, Sandlund JT, Jeha S, Pui CH, Howard SC. Clinical consequences of hyperglycemia during remission induction therapy for pediatric acute lymphoblastic leukemia. Leukemia. 2009 Feb;23(2):245-50. doi: 10.1038/leu.2008.289. Epub 2008 Oct 16. PMID 18923438
- [Background] French D, Yang W, Cheng C, Raimondi SC, Mullighan CG, Downing JR, Evans WE, Pui CH, Relling MV. Acquired variation outweighs inherited variation in whole genome analysis of methotrexate polyglutamate accumulation in leukemia. Blood. 2009 May 7;113(19):4512-20. doi: 10.1182/blood-2008-07-172106. Epub 2008 Dec 9. PMID 19066393
- [Background] Rubnitz JE, Onciu M, Pounds S, Shurtleff S, Cao X, Raimondi SC, Behm FG, Campana D, Razzouk BI, Ribeiro RC, Downing JR, Pui CH. Acute mixed lineage leukemia in children: the experience of St Jude Children's Research Hospital. Blood. 2009 May 21;113(21):5083-9. doi: 10.1182/blood-2008-10-187351. Epub 2009 Jan 8. PMID 19131545
- [Background] Pui CH, Campana D, Pei D, Bowman WP, Sandlund JT, Kaste SC, Ribeiro RC, Rubnitz JE, Raimondi SC, Onciu M, Coustan-Smith E, Kun LE, Jeha S, Cheng C, Howard SC, Simmons V, Bayles A, Metzger ML, Boyett JM, Leung W, Handgretinger R, Downing JR, Evans WE, Relling MV. Treating childhood acute lymphoblastic leukemia without cranial irradiation. N Engl J Med. 2009 Jun 25;360(26):2730-41. doi: 10.1056/NEJMoa0900386. PMID 19553647
- [Background] Mullighan CG, Collins-Underwood JR, Phillips LA, Loudin MG, Liu W, Zhang J, Ma J, Coustan-Smith E, Harvey RC, Willman CL, Mikhail FM, Meyer J, Carroll AJ, Williams RT, Cheng J, Heerema NA, Basso G, Pession A, Pui CH, Raimondi SC, Hunger SP, Downing JR, Carroll WL, Rabin KR. Rearrangement of CRLF2 in B-progenitor- and Down syndrome-associated acute lymphoblastic leukemia. Nat Genet. 2009 Nov;41(11):1243-6. doi: 10.1038/ng.469. Epub 2009 Oct 18. PMID 19838194
- [Background] Trevino LR, Shimasaki N, Yang W, Panetta JC, Cheng C, Pei D, Chan D, Sparreboom A, Giacomini KM, Pui CH, Evans WE, Relling MV. Germline genetic variation in an organic anion transporter polypeptide associated with methotrexate pharmacokinetics and clinical effects. J Clin Oncol. 2009 Dec 10;27(35):5972-8. doi: 10.1200/JCO.2008.20.4156. Epub 2009 Nov 9. PMID 19901119
- [Background] Spraker HL, Spyridis GP, Pui CH, Howard SC. Conservative management of pancreatic pseudocysts in children with acute lymphoblastic leukemia. J Pediatr Hematol Oncol. 2009 Dec;31(12):957-9. doi: 10.1097/MPH.0b013e3181ba9e6a. PMID 19956023
- [Background] Reddick WE, Glass JO, Johnson DP, Laningham FH, Pui CH. Voxel-based analysis of T2 hyperintensities in white matter during treatment of childhood leukemia. AJNR Am J Neuroradiol. 2009 Nov;30(10):1947-54. doi: 10.3174/ajnr.A1733. Epub 2009 Jul 30. PMID 19643920
- [Background] Stocco G, Cheok MH, Crews KR, Dervieux T, French D, Pei D, Yang W, Cheng C, Pui CH, Relling MV, Evans WE. Genetic polymorphism of inosine triphosphate pyrophosphatase is a determinant of mercaptopurine metabolism and toxicity during treatment for acute lymphoblastic leukemia. Clin Pharmacol Ther. 2009 Feb;85(2):164-72. doi: 10.1038/clpt.2008.154. Epub 2008 Aug 6. PMID 18685564
- [Background] Espinosa L, Cathelin S, D'Altri T, Trimarchi T, Statnikov A, Guiu J, Rodilla V, Ingles-Esteve J, Nomdedeu J, Bellosillo B, Besses C, Abdel-Wahab O, Kucine N, Sun SC, Song G, Mullighan CC, Levine RL, Rajewsky K, Aifantis I, Bigas A. The Notch/Hes1 pathway sustains NF-kappaB activation through CYLD repression in T cell leukemia. Cancer Cell. 2010 Sep 14;18(3):268-81. doi: 10.1016/j.ccr.2010.08.006. PMID 20832754
- [Background] Crews KR, Zhou Y, Pauley JL, Howard SC, Jeha S, Relling MV, Pui CH. Effect of allopurinol versus urate oxidase on methotrexate pharmacokinetics in children with newly diagnosed acute lymphoblastic leukemia. Cancer. 2010 Jan 1;116(1):227-32. doi: 10.1002/cncr.24681. PMID 19834958
- [Background] Yang W, Trevino LR, Yang JJ, Scheet P, Pui CH, Evans WE, Relling MV. ARID5B SNP rs10821936 is associated with risk of childhood acute lymphoblastic leukemia in blacks and contributes to racial differences in leukemia incidence. Leukemia. 2010 Apr;24(4):894-6. doi: 10.1038/leu.2009.277. Epub 2010 Jan 7. No abstract available. PMID 20054350
- [Background] Gutierrez A, Dahlberg SE, Neuberg DS, Zhang J, Grebliunaite R, Sanda T, Protopopov A, Tosello V, Kutok J, Larson RS, Borowitz MJ, Loh ML, Ferrando AA, Winter SS, Mullighan CG, Silverman LB, Chin L, Hunger SP, Sallan SE, Look AT. Absence of biallelic TCRgamma deletion predicts early treatment failure in pediatric T-cell acute lymphoblastic leukemia. J Clin Oncol. 2010 Aug 20;28(24):3816-23. doi: 10.1200/JCO.2010.28.3390. Epub 2010 Jul 19. PMID 20644084
- [Background] Stow P, Key L, Chen X, Pan Q, Neale GA, Coustan-Smith E, Mullighan CG, Zhou Y, Pui CH, Campana D. Clinical significance of low levels of minimal residual disease at the end of remission induction therapy in childhood acute lymphoblastic leukemia. Blood. 2010 Jun 10;115(23):4657-63. doi: 10.1182/blood-2009-11-253435. Epub 2010 Mar 19. PMID 20304809
- [Background] Panetta JC, Sparreboom A, Pui CH, Relling MV, Evans WE. Modeling mechanisms of in vivo variability in methotrexate accumulation and folate pathway inhibition in acute lymphoblastic leukemia cells. PLoS Comput Biol. 2010 Dec 2;6(12):e1001019. doi: 10.1371/journal.pcbi.1001019. PMID 21152005
- [Background] Campana D. Minimal residual disease in acute lymphoblastic leukemia. Hematology Am Soc Hematol Educ Program. 2010;2010:7-12. doi: 10.1182/asheducation-2010.1.7. PMID 21239764
- [Background] Caniza MA, Hunger SP, Schrauder A, Valsecchi MG, Pui CH, Masera G; Members of International Study Group of Childhood ALL ( "Ponte di Legno Working Group"). The controversy of varicella vaccination in children with acute lymphoblastic leukemia. Pediatr Blood Cancer. 2012 Jan;58(1):12-6. doi: 10.1002/pbc.22759. Epub 2010 Sep 16. PMID 20848637
- [Background] Ashford J, Schoffstall C, Reddick WE, Leone C, Laningham FH, Glass JO, Pei D, Cheng C, Pui CH, Conklin HM. Attention and working memory abilities in children treated for acute lymphoblastic leukemia. Cancer. 2010 Oct 1;116(19):4638-45. doi: 10.1002/cncr.25343. PMID 20572038
- [Background] Pui CH. Recent research advances in childhood acute lymphoblastic leukemia. J Formos Med Assoc. 2010 Nov;109(11):777-87. doi: 10.1016/S0929-6646(10)60123-4. PMID 21126650
- [Background] Anghelescu DL, Faughnan LG, Jeha S, Relling MV, Hinds PS, Sandlund JT, Cheng C, Pei D, Hankins G, Pauley JL, Pui CH. Neuropathic pain during treatment for childhood acute lymphoblastic leukemia. Pediatr Blood Cancer. 2011 Dec 15;57(7):1147-53. doi: 10.1002/pbc.23039. Epub 2011 Feb 11. PMID 21319291
- [Background] Pui CH, Pei D, Campana D, Bowman WP, Sandlund JT, Kaste SC, Ribeiro RC, Rubnitz JE, Coustan-Smith E, Jeha S, Cheng C, Metzger ML, Bhojwani D, Inaba H, Raimondi SC, Onciu M, Howard SC, Leung W, Downing JR, Evans WE, Relling MV. Improved prognosis for older adolescents with acute lymphoblastic leukemia. J Clin Oncol. 2011 Feb 1;29(4):386-91. doi: 10.1200/JCO.2010.32.0325. Epub 2010 Dec 20. PMID 21172890
- [Background] Rudner LA, Brown KH, Dobrinski KP, Bradley DF, Garcia MI, Smith AC, Downie JM, Meeker ND, Look AT, Downing JR, Gutierrez A, Mullighan CG, Schiffman JD, Lee C, Trede NS, Frazer JK. Shared acquired genomic changes in zebrafish and human T-ALL. Oncogene. 2011 Oct 13;30(41):4289-96. doi: 10.1038/onc.2011.138. Epub 2011 May 9. PMID 21552289
- [Background] Wang J, Mullighan CG, Easton J, Roberts S, Heatley SL, Ma J, Rusch MC, Chen K, Harris CC, Ding L, Holmfeldt L, Payne-Turner D, Fan X, Wei L, Zhao D, Obenauer JC, Naeve C, Mardis ER, Wilson RK, Downing JR, Zhang J. CREST maps somatic structural variation in cancer genomes with base-pair resolution. Nat Methods. 2011 Jun 12;8(8):652-4. doi: 10.1038/nmeth.1628. PMID 21666668
- [Background] Andersson AK, Miller DW, Lynch JA, Lemoff AS, Cai Z, Pounds SB, Radtke I, Yan B, Schuetz JD, Rubnitz JE, Ribeiro RC, Raimondi SC, Zhang J, Mullighan CG, Shurtleff SA, Schulman BA, Downing JR. IDH1 and IDH2 mutations in pediatric acute leukemia. Leukemia. 2011 Oct;25(10):1570-7. doi: 10.1038/leu.2011.133. Epub 2011 Jun 7. PMID 21647154
- [Background] Mullighan CG, Zhang J, Kasper LH, Lerach S, Payne-Turner D, Phillips LA, Heatley SL, Holmfeldt L, Collins-Underwood JR, Ma J, Buetow KH, Pui CH, Baker SD, Brindle PK, Downing JR. CREBBP mutations in relapsed acute lymphoblastic leukaemia. Nature. 2011 Mar 10;471(7337):235-9. doi: 10.1038/nature09727. PMID 21390130
- [Background] Kannan S, Fang W, Song G, Mullighan CG, Hammitt R, McMurray J, Zweidler-McKay PA. Notch/HES1-mediated PARP1 activation: a cell type-specific mechanism for tumor suppression. Blood. 2011 Mar 10;117(10):2891-900. doi: 10.1182/blood-2009-12-253419. Epub 2011 Jan 11. PMID 21224467
- [Background] Chen SH, Yang W, Fan Y, Stocco G, Crews KR, Yang JJ, Paugh SW, Pui CH, Evans WE, Relling MV. A genome-wide approach identifies that the aspartate metabolism pathway contributes to asparaginase sensitivity. Leukemia. 2011 Jan;25(1):66-74. doi: 10.1038/leu.2010.256. Epub 2010 Nov 12. PMID 21072045
- [Background] Crews KR, Cross SJ, McCormick JN, Baker DK, Molinelli AR, Mullins R, Relling MV, Hoffman JM. Development and implementation of a pharmacist-managed clinical pharmacogenetics service. Am J Health Syst Pharm. 2011 Jan 15;68(2):143-50. doi: 10.2146/ajhp100113. PMID 21200062
- [Background] Yang JJ, Cheng C, Devidas M, Cao X, Fan Y, Campana D, Yang W, Neale G, Cox NJ, Scheet P, Borowitz MJ, Winick NJ, Martin PL, Willman CL, Bowman WP, Camitta BM, Carroll A, Reaman GH, Carroll WL, Loh M, Hunger SP, Pui CH, Evans WE, Relling MV. Ancestry and pharmacogenomics of relapse in acute lymphoblastic leukemia. Nat Genet. 2011 Mar;43(3):237-41. doi: 10.1038/ng.763. Epub 2011 Feb 6. PMID 21297632
- [Background] Kim MJ, Skewes-Cox P, Fukushima H, Hesselson S, Yee SW, Ramsey LB, Nguyen L, Eshragh JL, Castro RA, Wen CC, Stryke D, Johns SJ, Ferrin TE, Kwok PY, Relling MV, Giacomini KM, Kroetz DL, Ahituv N. Functional characterization of liver enhancers that regulate drug-associated transporters. Clin Pharmacol Ther. 2011 Apr;89(4):571-8. doi: 10.1038/clpt.2010.353. Epub 2011 Mar 2. PMID 21368754
- [Background] Mikkelsen TS, Sparreboom A, Cheng C, Zhou Y, Boyett JM, Raimondi SC, Panetta JC, Bowman WP, Sandlund JT, Pui CH, Relling MV, Evans WE. Shortening infusion time for high-dose methotrexate alters antileukemic effects: a randomized prospective clinical trial. J Clin Oncol. 2011 May 1;29(13):1771-8. doi: 10.1200/JCO.2010.32.5340. Epub 2011 Mar 28. PMID 21444869
- [Background] Pounds S, Cao X, Cheng C, Yang JJ, Campana D, Pui CH, Evans WE, Relling MV. Integrated analysis of pharmacologic, clinical and SNP microarray data using Projection Onto the Most Interesting Statistical Evidence with Adaptive Permutation Testing. Int J Data Min Bioinform. 2011;5(2):143-57. doi: 10.1504/IJDMB.2011.039174. PMID 21516175
- [Background] Kawedia JD, Kaste SC, Pei D, Panetta JC, Cai X, Cheng C, Neale G, Howard SC, Evans WE, Pui CH, Relling MV. Pharmacokinetic, pharmacodynamic, and pharmacogenetic determinants of osteonecrosis in children with acute lymphoblastic leukemia. Blood. 2011 Feb 24;117(8):2340-7; quiz 2556. doi: 10.1182/blood-2010-10-311969. Epub 2010 Dec 10. PMID 21148812
- [Background] Coustan-Smith E, Song G, Clark C, Key L, Liu P, Mehrpooya M, Stow P, Su X, Shurtleff S, Pui CH, Downing JR, Campana D. New markers for minimal residual disease detection in acute lymphoblastic leukemia. Blood. 2011 Jun 9;117(23):6267-76. doi: 10.1182/blood-2010-12-324004. Epub 2011 Apr 12. PMID 21487112
- [Background] Leung W, Campana D, Yang J, Pei D, Coustan-Smith E, Gan K, Rubnitz JE, Sandlund JT, Ribeiro RC, Srinivasan A, Hartford C, Triplett BM, Dallas M, Pillai A, Handgretinger R, Laver JH, Pui CH. High success rate of hematopoietic cell transplantation regardless of donor source in children with very high-risk leukemia. Blood. 2011 Jul 14;118(2):223-30. doi: 10.1182/blood-2011-01-333070. Epub 2011 May 25. PMID 21613256
- [Background] Dumitrescu L, Brown-Gentry K, Goodloe R, Glenn K, Yang W, Kornegay N, Pui CH, Relling MV, Crawford DC. Evidence for age as a modifier of genetic associations for lipid levels. Ann Hum Genet. 2011 Sep;75(5):589-97. doi: 10.1111/j.1469-1809.2011.00664.x. Epub 2011 Jul 21. PMID 21777205
- [Background] Diouf B, Cheng Q, Krynetskaia NF, Yang W, Cheok M, Pei D, Fan Y, Cheng C, Krynetskiy EY, Geng H, Chen S, Thierfelder WE, Mullighan CG, Downing JR, Hsieh P, Pui CH, Relling MV, Evans WE. Somatic deletions of genes regulating MSH2 protein stability cause DNA mismatch repair deficiency and drug resistance in human leukemia cells. Nat Med. 2011 Sep 25;17(10):1298-303. doi: 10.1038/nm.2430. PMID 21946537
- [Background] Mikkelsen TS, Thorn CF, Yang JJ, Ulrich CM, French D, Zaza G, Dunnenberger HM, Marsh S, McLeod HL, Giacomini K, Becker ML, Gaedigk R, Leeder JS, Kager L, Relling MV, Evans W, Klein TE, Altman RB. PharmGKB summary: methotrexate pathway. Pharmacogenet Genomics. 2011 Oct;21(10):679-86. doi: 10.1097/FPC.0b013e328343dd93. No abstract available. PMID 21317831
- [Background] Krull KR, Khan RB, Ness KK, Ledet D, Zhu L, Pui CH, Howard SC, Srivastava DK, Sabin ND, Hudson MM, Morris EB. Symptoms of attention-deficit/hyperactivity disorder in long-term survivors of childhood leukemia. Pediatr Blood Cancer. 2011 Dec 15;57(7):1191-6. doi: 10.1002/pbc.22994. Epub 2011 Jan 28. PMID 21280202
- [Background] Zhang J, Ding L, Holmfeldt L, Wu G, Heatley SL, Payne-Turner D, Easton J, Chen X, Wang J, Rusch M, Lu C, Chen SC, Wei L, Collins-Underwood JR, Ma J, Roberts KG, Pounds SB, Ulyanov A, Becksfort J, Gupta P, Huether R, Kriwacki RW, Parker M, McGoldrick DJ, Zhao D, Alford D, Espy S, Bobba KC, Song G, Pei D, Cheng C, Roberts S, Barbato MI, Campana D, Coustan-Smith E, Shurtleff SA, Raimondi SC, Kleppe M, Cools J, Shimano KA, Hermiston ML, Doulatov S, Eppert K, Laurenti E, Notta F, Dick JE, Basso G, Hunger SP, Loh ML, Devidas M, Wood B, Winter S, Dunsmore KP, Fulton RS, Fulton LL, Hong X, Harris CC, Dooling DJ, Ochoa K, Johnson KJ, Obenauer JC, Evans WE, Pui CH, Naeve CW, Ley TJ, Mardis ER, Wilson RK, Downing JR, Mullighan CG. The genetic basis of early T-cell precursor acute lymphoblastic leukaemia. Nature. 2012 Jan 11;481(7380):157-63. doi: 10.1038/nature10725. PMID 22237106
- [Background] Christensen AM, Pauley JL, Molinelli AR, Panetta JC, Ward DA, Stewart CF, Hoffman JM, Howard SC, Pui CH, Pappo AS, Relling MV, Crews KR. Resumption of high-dose methotrexate after acute kidney injury and glucarpidase use in pediatric oncology patients. Cancer. 2012 Sep 1;118(17):4321-30. doi: 10.1002/cncr.27378. Epub 2012 Jan 17. PMID 22252903
- [Background] Bhojwani D, Pei D, Sandlund JT, Jeha S, Ribeiro RC, Rubnitz JE, Raimondi SC, Shurtleff S, Onciu M, Cheng C, Coustan-Smith E, Bowman WP, Howard SC, Metzger ML, Inaba H, Leung W, Evans WE, Campana D, Relling MV, Pui CH. ETV6-RUNX1-positive childhood acute lymphoblastic leukemia: improved outcome with contemporary therapy. Leukemia. 2012 Feb;26(2):265-70. doi: 10.1038/leu.2011.227. Epub 2011 Aug 26. PMID 21869842
- [Background] Kawedia JD, Liu C, Pei D, Cheng C, Fernandez CA, Howard SC, Campana D, Panetta JC, Bowman WP, Evans WE, Pui CH, Relling MV. Dexamethasone exposure and asparaginase antibodies affect relapse risk in acute lymphoblastic leukemia. Blood. 2012 Feb 16;119(7):1658-64. doi: 10.1182/blood-2011-09-381731. Epub 2011 Nov 23. PMID 22117041
- [Background] Ciarimboli G, Lancaster CS, Schlatter E, Franke RM, Sprowl JA, Pavenstadt H, Massmann V, Guckel D, Mathijssen RH, Yang W, Pui CH, Relling MV, Herrmann E, Sparreboom A. Proximal tubular secretion of creatinine by organic cation transporter OCT2 in cancer patients. Clin Cancer Res. 2012 Feb 15;18(4):1101-8. doi: 10.1158/1078-0432.CCR-11-2503. Epub 2012 Jan 5. PMID 22223530
- [Background] Xu H, Cheng C, Devidas M, Pei D, Fan Y, Yang W, Neale G, Scheet P, Burchard EG, Torgerson DG, Eng C, Dean M, Antillon F, Winick NJ, Martin PL, Willman CL, Camitta BM, Reaman GH, Carroll WL, Loh M, Evans WE, Pui CH, Hunger SP, Relling MV, Yang JJ. ARID5B genetic polymorphisms contribute to racial disparities in the incidence and treatment outcome of childhood acute lymphoblastic leukemia. J Clin Oncol. 2012 Mar 1;30(7):751-7. doi: 10.1200/JCO.2011.38.0345. Epub 2012 Jan 30. PMID 22291082
- [Background] Liu C, Kawedia JD, Cheng C, Pei D, Fernandez CA, Cai X, Crews KR, Kaste SC, Panetta JC, Bowman WP, Jeha S, Sandlund JT, Evans WE, Pui CH, Relling MV. Clinical utility and implications of asparaginase antibodies in acute lymphoblastic leukemia. Leukemia. 2012 Nov;26(11):2303-9. doi: 10.1038/leu.2012.102. Epub 2012 Apr 9. PMID 22484422
- [Background] Pui CH, Pei D, Pappo AS, Howard SC, Cheng C, Sandlund JT, Furman WL, Ribeiro RC, Spunt SL, Rubnitz JE, Jeha S, Hudson MM, Kun LE, Merchant TE, Kocak M, Broniscer A, Metzger ML, Downing JR, Leung W, Evans WE, Gajjar A. Treatment outcomes in black and white children with cancer: results from the SEER database and St Jude Children's Research Hospital, 1992 through 2007. J Clin Oncol. 2012 Jun 1;30(16):2005-12. doi: 10.1200/JCO.2011.40.8617. Epub 2012 Apr 30. PMID 22547602
- [Background] Ramsey LB, Bruun GH, Yang W, Trevino LR, Vattathil S, Scheet P, Cheng C, Rosner GL, Giacomini KM, Fan Y, Sparreboom A, Mikkelsen TS, Corydon TJ, Pui CH, Evans WE, Relling MV. Rare versus common variants in pharmacogenetics: SLCO1B1 variation and methotrexate disposition. Genome Res. 2012 Jan;22(1):1-8. doi: 10.1101/gr.129668.111. Epub 2011 Dec 6. PMID 22147369
- [Background] Leung W, Pui CH, Coustan-Smith E, Yang J, Pei D, Gan K, Srinivasan A, Hartford C, Triplett BM, Dallas M, Pillai A, Shook D, Rubnitz JE, Sandlund JT, Jeha S, Inaba H, Ribeiro RC, Handgretinger R, Laver JH, Campana D. Detectable minimal residual disease before hematopoietic cell transplantation is prognostic but does not preclude cure for children with very-high-risk leukemia. Blood. 2012 Jul 12;120(2):468-72. doi: 10.1182/blood-2012-02-409813. Epub 2012 Apr 19. PMID 22517895
- [Background] Pui CH, Mullighan CG, Evans WE, Relling MV. Pediatric acute lymphoblastic leukemia: where are we going and how do we get there? Blood. 2012 Aug 9;120(6):1165-74. doi: 10.1182/blood-2012-05-378943. Epub 2012 Jun 22. PMID 22730540
- [Background] Roberts KG, Morin RD, Zhang J, Hirst M, Zhao Y, Su X, Chen SC, Payne-Turner D, Churchman ML, Harvey RC, Chen X, Kasap C, Yan C, Becksfort J, Finney RP, Teachey DT, Maude SL, Tse K, Moore R, Jones S, Mungall K, Birol I, Edmonson MN, Hu Y, Buetow KE, Chen IM, Carroll WL, Wei L, Ma J, Kleppe M, Levine RL, Garcia-Manero G, Larsen E, Shah NP, Devidas M, Reaman G, Smith M, Paugh SW, Evans WE, Grupp SA, Jeha S, Pui CH, Gerhard DS, Downing JR, Willman CL, Loh M, Hunger SP, Marra MA, Mullighan CG. Genetic alterations activating kinase and cytokine receptor signaling in high-risk acute lymphoblastic leukemia. Cancer Cell. 2012 Aug 14;22(2):153-66. doi: 10.1016/j.ccr.2012.06.005. PMID 22897847
- [Background] Conklin HM, Krull KR, Reddick WE, Pei D, Cheng C, Pui CH. Cognitive outcomes following contemporary treatment without cranial irradiation for childhood acute lymphoblastic leukemia. J Natl Cancer Inst. 2012 Sep 19;104(18):1386-95. doi: 10.1093/jnci/djs344. Epub 2012 Aug 27. PMID 22927505
- [Background] Stocco G, Yang W, Crews KR, Thierfelder WE, Decorti G, Londero M, Franca R, Rabusin M, Valsecchi MG, Pei D, Cheng C, Paugh SW, Ramsey LB, Diouf B, McCorkle JR, Jones TS, Pui CH, Relling MV, Evans WE. PACSIN2 polymorphism influences TPMT activity and mercaptopurine-related gastrointestinal toxicity. Hum Mol Genet. 2012 Nov 1;21(21):4793-804. doi: 10.1093/hmg/dds302. Epub 2012 Jul 30. PMID 22846425
- [Background] Yang JJ, Cheng C, Devidas M, Cao X, Campana D, Yang W, Fan Y, Neale G, Cox N, Scheet P, Borowitz MJ, Winick NJ, Martin PL, Bowman WP, Camitta B, Reaman GH, Carroll WL, Willman CL, Hunger SP, Evans WE, Pui CH, Loh M, Relling MV. Genome-wide association study identifies germline polymorphisms associated with relapse of childhood acute lymphoblastic leukemia. Blood. 2012 Nov 15;120(20):4197-204. doi: 10.1182/blood-2012-07-440107. Epub 2012 Sep 24. PMID 23007406
- [Background] Anghelescu DL, Burgoyne LL, Faughnan LG, Hankins GM, Smeltzer MP, Pui CH. Prospective randomized crossover evaluation of three anesthetic regimens for painful procedures in children with cancer. J Pediatr. 2013 Jan;162(1):137-41. doi: 10.1016/j.jpeds.2012.06.056. Epub 2012 Aug 9. PMID 22883421
- [Background] Ramsey LB, Panetta JC, Smith C, Yang W, Fan Y, Winick NJ, Martin PL, Cheng C, Devidas M, Pui CH, Evans WE, Hunger SP, Loh M, Relling MV. Genome-wide study of methotrexate clearance replicates SLCO1B1. Blood. 2013 Feb 7;121(6):898-904. doi: 10.1182/blood-2012-08-452839. Epub 2012 Dec 11. PMID 23233662
- [Background] Holmfeldt L, Wei L, Diaz-Flores E, Walsh M, Zhang J, Ding L, Payne-Turner D, Churchman M, Andersson A, Chen SC, McCastlain K, Becksfort J, Ma J, Wu G, Patel SN, Heatley SL, Phillips LA, Song G, Easton J, Parker M, Chen X, Rusch M, Boggs K, Vadodaria B, Hedlund E, Drenberg C, Baker S, Pei D, Cheng C, Huether R, Lu C, Fulton RS, Fulton LL, Tabib Y, Dooling DJ, Ochoa K, Minden M, Lewis ID, To LB, Marlton P, Roberts AW, Raca G, Stock W, Neale G, Drexler HG, Dickins RA, Ellison DW, Shurtleff SA, Pui CH, Ribeiro RC, Devidas M, Carroll AJ, Heerema NA, Wood B, Borowitz MJ, Gastier-Foster JM, Raimondi SC, Mardis ER, Wilson RK, Downing JR, Hunger SP, Loh ML, Mullighan CG. The genomic landscape of hypodiploid acute lymphoblastic leukemia. Nat Genet. 2013 Mar;45(3):242-52. doi: 10.1038/ng.2532. Epub 2013 Jan 20. PMID 23334668
- [Background] Xu H, Yang W, Perez-Andreu V, Devidas M, Fan Y, Cheng C, Pei D, Scheet P, Burchard EG, Eng C, Huntsman S, Torgerson DG, Dean M, Winick NJ, Martin PL, Camitta BM, Bowman WP, Willman CL, Carroll WL, Mullighan CG, Bhojwani D, Hunger SP, Pui CH, Evans WE, Relling MV, Loh ML, Yang JJ. Novel susceptibility variants at 10p12.31-12.2 for childhood acute lymphoblastic leukemia in ethnically diverse populations. J Natl Cancer Inst. 2013 May 15;105(10):733-42. doi: 10.1093/jnci/djt042. Epub 2013 Mar 19. PMID 23512250
- [Background] Krull KR, Bhojwani D, Conklin HM, Pei D, Cheng C, Reddick WE, Sandlund JT, Pui CH. Genetic mediators of neurocognitive outcomes in survivors of childhood acute lymphoblastic leukemia. J Clin Oncol. 2013 Jun 10;31(17):2182-8. doi: 10.1200/JCO.2012.46.7944. Epub 2013 May 6. PMID 23650422
- [Background] Pauley JL, Panetta JC, Crews KR, Pei D, Cheng C, McCormick J, Howard SC, Sandlund JT, Jeha S, Ribeiro R, Rubnitz J, Pui CH, Evans WE, Relling MV. Between-course targeting of methotrexate exposure using pharmacokinetically guided dosage adjustments. Cancer Chemother Pharmacol. 2013 Aug;72(2):369-78. doi: 10.1007/s00280-013-2206-x. Epub 2013 Jun 13. PMID 23760811
- [Background] Rubnitz JE, Campbell P, Zhou Y, Sandlund JT, Jeha S, Ribeiro RC, Inaba H, Bhojwani D, Relling MV, Howard SC, Campana D, Pui CH. Prognostic impact of absolute lymphocyte counts at the end of remission induction in childhood acute lymphoblastic leukemia. Cancer. 2013 Jun 1;119(11):2061-6. doi: 10.1002/cncr.28026. Epub 2013 Mar 1. PMID 23456849
- [Background] Wright KD, Onciu MM, Coustan-Smith E, Campana D, Raimondi SC, Inaba H, Ribeiro R, Pui CH, Sandlund JT. Successful treatment of pediatric plasmacytoid dendritic cell tumors with a contemporary regimen for acute lymphoblastic leukemia. Pediatr Blood Cancer. 2013 Jul;60(7):E38-41. doi: 10.1002/pbc.24483. Epub 2013 Feb 15. PMID 23417921
- [Background] Jeha S, Coustan-Smith E, Pei D, Sandlund JT, Rubnitz JE, Howard SC, Inaba H, Bhojwani D, Metzger ML, Cheng C, Choi JK, Jacobsen J, Shurtleff SA, Raimondi S, Ribeiro RC, Pui CH, Campana D. Impact of tyrosine kinase inhibitors on minimal residual disease and outcome in childhood Philadelphia chromosome-positive acute lymphoblastic leukemia. Cancer. 2014 May 15;120(10):1514-9. doi: 10.1002/cncr.28598. Epub 2014 Feb 5. PMID 24501014
- [Background] Bhojwani D, Sabin ND, Pei D, Yang JJ, Khan RB, Panetta JC, Krull KR, Inaba H, Rubnitz JE, Metzger ML, Howard SC, Ribeiro RC, Cheng C, Reddick WE, Jeha S, Sandlund JT, Evans WE, Pui CH, Relling MV. Methotrexate-induced neurotoxicity and leukoencephalopathy in childhood acute lymphoblastic leukemia. J Clin Oncol. 2014 Mar 20;32(9):949-59. doi: 10.1200/JCO.2013.53.0808. Epub 2014 Feb 18. PMID 24550419
- [Background] Pui CH, Pei D, Campana D, Cheng C, Sandlund JT, Bowman WP, Hudson MM, Ribeiro RC, Raimondi SC, Jeha S, Howard SC, Bhojwani D, Inaba H, Rubnitz JE, Metzger ML, Gruber TA, Coustan-Smith E, Downing JR, Leung WH, Relling MV, Evans WE. A revised definition for cure of childhood acute lymphoblastic leukemia. Leukemia. 2014 Dec;28(12):2336-43. doi: 10.1038/leu.2014.142. Epub 2014 Apr 30. PMID 24781017
- [Background] Roberts KG, Pei D, Campana D, Payne-Turner D, Li Y, Cheng C, Sandlund JT, Jeha S, Easton J, Becksfort J, Zhang J, Coustan-Smith E, Raimondi SC, Leung WH, Relling MV, Evans WE, Downing JR, Mullighan CG, Pui CH. Outcomes of children with BCR-ABL1-like acute lymphoblastic leukemia treated with risk-directed therapy based on the levels of minimal residual disease. J Clin Oncol. 2014 Sep 20;32(27):3012-20. doi: 10.1200/JCO.2014.55.4105. PMID 25049327
- [Background] Pui CH, Evans WE. A 50-year journey to cure childhood acute lymphoblastic leukemia. Semin Hematol. 2013 Jul;50(3):185-96. doi: 10.1053/j.seminhematol.2013.06.007. PMID 23953334
- [Background] Perez-Andreu V, Roberts KG, Harvey RC, Yang W, Cheng C, Pei D, Xu H, Gastier-Foster J, E S, Lim JY, Chen IM, Fan Y, Devidas M, Borowitz MJ, Smith C, Neale G, Burchard EG, Torgerson DG, Klussmann FA, Villagran CR, Winick NJ, Camitta BM, Raetz E, Wood B, Yue F, Carroll WL, Larsen E, Bowman WP, Loh ML, Dean M, Bhojwani D, Pui CH, Evans WE, Relling MV, Hunger SP, Willman CL, Mullighan CG, Yang JJ. Inherited GATA3 variants are associated with Ph-like childhood acute lymphoblastic leukemia and risk of relapse. Nat Genet. 2013 Dec;45(12):1494-8. doi: 10.1038/ng.2803. Epub 2013 Oct 20. PMID 24141364
- [Background] Krull KR, Brinkman TM, Li C, Armstrong GT, Ness KK, Srivastava DK, Gurney JG, Kimberg C, Krasin MJ, Pui CH, Robison LL, Hudson MM. Neurocognitive outcomes decades after treatment for childhood acute lymphoblastic leukemia: a report from the St Jude lifetime cohort study. J Clin Oncol. 2013 Dec 10;31(35):4407-15. doi: 10.1200/JCO.2012.48.2315. Epub 2013 Nov 4. PMID 24190124
- [Background] Kaste SC, Qi A, Smith K, Surprise H, Lovorn E, Boyett J, Ferry RJ Jr, Relling MV, Shurtleff SA, Pui CH, Carbone L, Hudson MM, Ness KK. Calcium and cholecalciferol supplementation provides no added benefit to nutritional counseling to improve bone mineral density in survivors of childhood acute lymphoblastic leukemia (ALL). Pediatr Blood Cancer. 2014 May;61(5):885-93. doi: 10.1002/pbc.24882. Epub 2014 Jan 7. PMID 24395288
- [Background] Esbenshade AJ, Friedman DL, Smith WA, Jeha S, Pui CH, Robison LL, Ness KK. Feasibility and initial effectiveness of home exercise during maintenance therapy for childhood acute lymphoblastic leukemia. Pediatr Phys Ther. 2014 Fall;26(3):301-7. doi: 10.1097/PEP.0000000000000053. PMID 24979081
- [Background] Watsky MA, Carbone LD, An Q, Cheng C, Lovorn EA, Hudson MM, Pui CH, Kaste SC. Bone turnover in long-term survivors of childhood acute lymphoblastic leukemia. Pediatr Blood Cancer. 2014 Aug;61(8):1451-6. doi: 10.1002/pbc.25025. Epub 2014 Mar 20. PMID 24648266
- [Background] Fernandez CA, Smith C, Yang W, Date M, Bashford D, Larsen E, Bowman WP, Liu C, Ramsey LB, Chang T, Turner V, Loh ML, Raetz EA, Winick NJ, Hunger SP, Carroll WL, Onengut-Gumuscu S, Chen WM, Concannon P, Rich SS, Scheet P, Jeha S, Pui CH, Evans WE, Devidas M, Relling MV. HLA-DRB1*07:01 is associated with a higher risk of asparaginase allergies. Blood. 2014 Aug 21;124(8):1266-76. doi: 10.1182/blood-2014-03-563742. Epub 2014 Jun 26. PMID 24970932
- [Background] Khan RB, Hudson MM, Ledet DS, Morris EB, Pui CH, Howard SC, Krull KR, Hinds PS, Crom D, Browne E, Zhu L, Rai S, Srivastava D, Ness KK. Neurologic morbidity and quality of life in survivors of childhood acute lymphoblastic leukemia: a prospective cross-sectional study. J Cancer Surviv. 2014 Dec;8(4):688-96. doi: 10.1007/s11764-014-0375-1. Epub 2014 Jul 10. PMID 25008582
- [Background] Sadighi ZS, Ness KK, Hudson MM, Morris EB, Ledet DS, Pui CH, Howard SC, Krull KR, Browne E, Crom D, Hinds PS, Zhu L, Srivastava D, Khan RB. Headache types, related morbidity, and quality of life in survivors of childhood acute lymphoblastic leukemia: a prospective cross sectional study. Eur J Paediatr Neurol. 2014 Nov;18(6):722-9. doi: 10.1016/j.ejpn.2014.06.006. Epub 2014 Jul 5. PMID 25030329
- [Background] Bhojwani D, Darbandi R, Pei D, Ramsey LB, Chemaitilly W, Sandlund JT, Cheng C, Pui CH, Relling MV, Jeha S, Metzger ML. Severe hypertriglyceridaemia during therapy for childhood acute lymphoblastic leukaemia. Eur J Cancer. 2014 Oct;50(15):2685-94. doi: 10.1016/j.ejca.2014.06.023. Epub 2014 Jul 30. PMID 25087182
- [Background] Roberts KG, Li Y, Payne-Turner D, Harvey RC, Yang YL, Pei D, McCastlain K, Ding L, Lu C, Song G, Ma J, Becksfort J, Rusch M, Chen SC, Easton J, Cheng J, Boggs K, Santiago-Morales N, Iacobucci I, Fulton RS, Wen J, Valentine M, Cheng C, Paugh SW, Devidas M, Chen IM, Reshmi S, Smith A, Hedlund E, Gupta P, Nagahawatte P, Wu G, Chen X, Yergeau D, Vadodaria B, Mulder H, Winick NJ, Larsen EC, Carroll WL, Heerema NA, Carroll AJ, Grayson G, Tasian SK, Moore AS, Keller F, Frei-Jones M, Whitlock JA, Raetz EA, White DL, Hughes TP, Guidry Auvil JM, Smith MA, Marcucci G, Bloomfield CD, Mrozek K, Kohlschmidt J, Stock W, Kornblau SM, Konopleva M, Paietta E, Pui CH, Jeha S, Relling MV, Evans WE, Gerhard DS, Gastier-Foster JM, Mardis E, Wilson RK, Loh ML, Downing JR, Hunger SP, Willman CL, Zhang J, Mullighan CG. Targetable kinase-activating lesions in Ph-like acute lymphoblastic leukemia. N Engl J Med. 2014 Sep 11;371(11):1005-15. doi: 10.1056/NEJMoa1403088. PMID 25207766
- [Background] Sullivan EM, Jeha S, Kang G, Cheng C, Rooney B, Holladay M, Bari R, Schell S, Tuggle M, Pui CH, Leung W. NK cell genotype and phenotype at diagnosis of acute lymphoblastic leukemia correlate with postinduction residual disease. Clin Cancer Res. 2014 Dec 1;20(23):5986-94. doi: 10.1158/1078-0432.CCR-14-0479. Epub 2014 Oct 3. PMID 25281696
- [Background] Ness KK, Kaste SC, Zhu L, Pui CH, Jeha S, Nathan PC, Inaba H, Wasilewski-Masker K, Shah D, Wells RJ, Karlage RE, Robison LL, Cox CL. Skeletal, neuromuscular and fitness impairments among children with newly diagnosed acute lymphoblastic leukemia. Leuk Lymphoma. 2015 Apr;56(4):1004-11. doi: 10.3109/10428194.2014.944519. Epub 2014 Aug 20. PMID 25030039
- [Background] Perez-Andreu V, Roberts KG, Xu H, Smith C, Zhang H, Yang W, Harvey RC, Payne-Turner D, Devidas M, Cheng IM, Carroll WL, Heerema NA, Carroll AJ, Raetz EA, Gastier-Foster JM, Marcucci G, Bloomfield CD, Mrozek K, Kohlschmidt J, Stock W, Kornblau SM, Konopleva M, Paietta E, Rowe JM, Luger SM, Tallman MS, Dean M, Burchard EG, Torgerson DG, Yue F, Wang Y, Pui CH, Jeha S, Relling MV, Evans WE, Gerhard DS, Loh ML, Willman CL, Hunger SP, Mullighan CG, Yang JJ. A genome-wide association study of susceptibility to acute lymphoblastic leukemia in adolescents and young adults. Blood. 2015 Jan 22;125(4):680-6. doi: 10.1182/blood-2014-09-595744. Epub 2014 Dec 2. PMID 25468567
- [Background] Fernandez CA, Smith C, Karol SE, Ramsey LB, Liu C, Pui CH, Jeha S, Evans WE, Finkelman FD, Relling MV. Effect of premedications in a murine model of asparaginase hypersensitivity. J Pharmacol Exp Ther. 2015 Mar;352(3):541-51. doi: 10.1124/jpet.114.220780. Epub 2015 Jan 8. PMID 25573198
- [Background] Malpert AV, Kimberg C, Luxton J, Mullins LL, Pui CH, Hudson MM, Krull KR, Brinkman TM. Emotional distress in parents of long-term survivors of childhood acute lymphoblastic leukemia. Psychooncology. 2015 Sep;24(9):1116-23. doi: 10.1002/pon.3732. Epub 2014 Dec 29. PMID 25557175
- [Background] Kaste SC, Pei D, Cheng C, Neel MD, Bowman WP, Ribeiro RC, Metzger ML, Bhojwani D, Inaba H, Campbell P, Rubnitz JE, Jeha S, Sandlund JT, Downing JR, Relling MV, Pui CH, Howard SC. Utility of early screening magnetic resonance imaging for extensive hip osteonecrosis in pediatric patients treated with glucocorticoids. J Clin Oncol. 2015 Feb 20;33(6):610-5. doi: 10.1200/JCO.2014.57.5480. Epub 2015 Jan 20. PMID 25605853
- [Background] Yang JJ, Landier W, Yang W, Liu C, Hageman L, Cheng C, Pei D, Chen Y, Crews KR, Kornegay N, Wong FL, Evans WE, Pui CH, Bhatia S, Relling MV. Inherited NUDT15 variant is a genetic determinant of mercaptopurine intolerance in children with acute lymphoblastic leukemia. J Clin Oncol. 2015 Apr 10;33(11):1235-42. doi: 10.1200/JCO.2014.59.4671. Epub 2015 Jan 26. PMID 25624441
- [Background] Diouf B, Crews KR, Lew G, Pei D, Cheng C, Bao J, Zheng JJ, Yang W, Fan Y, Wheeler HE, Wing C, Delaney SM, Komatsu M, Paugh SW, McCorkle JR, Lu X, Winick NJ, Carroll WL, Loh ML, Hunger SP, Devidas M, Pui CH, Dolan ME, Relling MV, Evans WE. Association of an inherited genetic variant with vincristine-related peripheral neuropathy in children with acute lymphoblastic leukemia. JAMA. 2015 Feb 24;313(8):815-23. doi: 10.1001/jama.2015.0894. PMID 25710658
- [Background] Andersson AK, Ma J, Wang J, Chen X, Gedman AL, Dang J, Nakitandwe J, Holmfeldt L, Parker M, Easton J, Huether R, Kriwacki R, Rusch M, Wu G, Li Y, Mulder H, Raimondi S, Pounds S, Kang G, Shi L, Becksfort J, Gupta P, Payne-Turner D, Vadodaria B, Boggs K, Yergeau D, Manne J, Song G, Edmonson M, Nagahawatte P, Wei L, Cheng C, Pei D, Sutton R, Venn NC, Chetcuti A, Rush A, Catchpoole D, Heldrup J, Fioretos T, Lu C, Ding L, Pui CH, Shurtleff S, Mullighan CG, Mardis ER, Wilson RK, Gruber TA, Zhang J, Downing JR; St. Jude Children's Research Hospital-Washington University Pediatric Cancer Genome Project. The landscape of somatic mutations in infant MLL-rearranged acute lymphoblastic leukemias. Nat Genet. 2015 Apr;47(4):330-7. doi: 10.1038/ng.3230. Epub 2015 Mar 2. PMID 25730765
- [Background] Pui CH, Pei D, Coustan-Smith E, Jeha S, Cheng C, Bowman WP, Sandlund JT, Ribeiro RC, Rubnitz JE, Inaba H, Bhojwani D, Gruber TA, Leung WH, Downing JR, Evans WE, Relling MV, Campana D. Clinical utility of sequential minimal residual disease measurements in the context of risk-based therapy in childhood acute lymphoblastic leukaemia: a prospective study. Lancet Oncol. 2015 Apr;16(4):465-74. doi: 10.1016/S1470-2045(15)70082-3. Epub 2015 Mar 20. PMID 25800893
- [Background] Ness KK, DeLany JP, Kaste SC, Mulrooney DA, Pui CH, Chemaitilly W, Karlage RE, Lanctot JQ, Howell CR, Lu L, Srivastava DK, Robison LL, Hudson MM. Energy balance and fitness in adult survivors of childhood acute lymphoblastic leukemia. Blood. 2015 May 28;125(22):3411-9. doi: 10.1182/blood-2015-01-621680. Epub 2015 Mar 26. PMID 25814529
- [Background] Paugh SW, Bonten EJ, Savic D, Ramsey LB, Thierfelder WE, Gurung P, Malireddi RK, Actis M, Mayasundari A, Min J, Coss DR, Laudermilk LT, Panetta JC, McCorkle JR, Fan Y, Crews KR, Stocco G, Wilkinson MR, Ferreira AM, Cheng C, Yang W, Karol SE, Fernandez CA, Diouf B, Smith C, Hicks JK, Zanut A, Giordanengo A, Crona D, Bianchi JJ, Holmfeldt L, Mullighan CG, den Boer ML, Pieters R, Jeha S, Dunwell TL, Latif F, Bhojwani D, Carroll WL, Pui CH, Myers RM, Guy RK, Kanneganti TD, Relling MV, Evans WE. NALP3 inflammasome upregulation and CASP1 cleavage of the glucocorticoid receptor cause glucocorticoid resistance in leukemia cells. Nat Genet. 2015 Jun;47(6):607-14. doi: 10.1038/ng.3283. Epub 2015 May 4. PMID 25938942
- [Background] Bi W, Kang G, Zhao Y, Cui Y, Yan S, Li Y, Cheng C, Pounds SB, Borowitz MJ, Relling MV, Yang JJ, Liu Z, Pui CH, Hunger SP, Hartford CM, Leung W, Zhang JF. SVSI: fast and powerful set-valued system identification approach to identifying rare variants in sequencing studies for ordered categorical traits. Ann Hum Genet. 2015 Jul;79(4):294-309. doi: 10.1111/ahg.12117. Epub 2015 May 11. PMID 25959545
- [Background] Fernandez CA, Smith C, Yang W, Mullighan CG, Qu C, Larsen E, Bowman WP, Liu C, Ramsey LB, Chang T, Karol SE, Loh ML, Raetz EA, Winick NJ, Hunger SP, Carroll WL, Jeha S, Pui CH, Evans WE, Devidas M, Relling MV. Genome-wide analysis links NFATC2 with asparaginase hypersensitivity. Blood. 2015 Jul 2;126(1):69-75. doi: 10.1182/blood-2015-02-628800. Epub 2015 May 18. PMID 25987655
- [Background] Pui CH, Yang JJ, Hunger SP, Pieters R, Schrappe M, Biondi A, Vora A, Baruchel A, Silverman LB, Schmiegelow K, Escherich G, Horibe K, Benoit YC, Izraeli S, Yeoh AE, Liang DC, Downing JR, Evans WE, Relling MV, Mullighan CG. Childhood Acute Lymphoblastic Leukemia: Progress Through Collaboration. J Clin Oncol. 2015 Sep 20;33(27):2938-48. doi: 10.1200/JCO.2014.59.1636. Epub 2015 Aug 24. PMID 26304874
- [Background] Xu H, Zhang H, Yang W, Yadav R, Morrison AC, Qian M, Devidas M, Liu Y, Perez-Andreu V, Zhao X, Gastier-Foster JM, Lupo PJ, Neale G, Raetz E, Larsen E, Bowman WP, Carroll WL, Winick N, Williams R, Hansen T, Holm JC, Mardis E, Fulton R, Pui CH, Zhang J, Mullighan CG, Evans WE, Hunger SP, Gupta R, Schmiegelow K, Loh ML, Relling MV, Yang JJ. Inherited coding variants at the CDKN2A locus influence susceptibility to acute lymphoblastic leukaemia in children. Nat Commun. 2015 Jun 24;6:7553. doi: 10.1038/ncomms8553. PMID 26104880
- [Background] Topka S, Vijai J, Walsh MF, Jacobs L, Maria A, Villano D, Gaddam P, Wu G, McGee RB, Quinn E, Inaba H, Hartford C, Pui CH, Pappo A, Edmonson M, Zhang MY, Stepensky P, Steinherz P, Schrader K, Lincoln A, Bussel J, Lipkin SM, Goldgur Y, Harit M, Stadler ZK, Mullighan C, Weintraub M, Shimamura A, Zhang J, Downing JR, Nichols KE, Offit K. Germline ETV6 Mutations Confer Susceptibility to Acute Lymphoblastic Leukemia and Thrombocytopenia. PLoS Genet. 2015 Jun 23;11(6):e1005262. doi: 10.1371/journal.pgen.1005262. eCollection 2015 Jun. PMID 26102509
- [Background] Bari R, Hartford C, Chan WK, Vong Q, Li Y, Gan K, Zhou Y, Cheng C, Kang G, Shurtleff S, Turner V, Pui CH, Downing JR, Leung W. Genome-wide single-nucleotide polymorphism analysis revealed SUFU suppression of acute graft-versus-host disease through downregulation of HLA-DR expression in recipient dendritic cells. Sci Rep. 2015 Jun 11;5:11098. doi: 10.1038/srep11098. PMID 26067905
- [Background] Ramsey LB, Janke LJ, Payton MA, Cai X, Paugh SW, Karol SE, Kamdem Kamdem L, Cheng C, Williams RT, Jeha S, Pui CH, Evans WE, Relling MV. Antileukemic Efficacy of Continuous vs Discontinuous Dexamethasone in Murine Models of Acute Lymphoblastic Leukemia. PLoS One. 2015 Aug 7;10(8):e0135134. doi: 10.1371/journal.pone.0135134. eCollection 2015. PMID 26252865
- [Background] Karol SE, Yang W, Van Driest SL, Chang TY, Kaste S, Bowton E, Basford M, Bastarache L, Roden DM, Denny JC, Larsen E, Winick N, Carroll WL, Cheng C, Pei D, Fernandez CA, Liu C, Smith C, Loh ML, Raetz EA, Hunger SP, Scheet P, Jeha S, Pui CH, Evans WE, Devidas M, Mattano LA Jr, Relling MV. Genetics of glucocorticoid-associated osteonecrosis in children with acute lymphoblastic leukemia. Blood. 2015 Oct 8;126(15):1770-6. doi: 10.1182/blood-2015-05-643601. Epub 2015 Aug 11. PMID 26265699
- [Background] Zhang J, Walsh MF, Wu G, Edmonson MN, Gruber TA, Easton J, Hedges D, Ma X, Zhou X, Yergeau DA, Wilkinson MR, Vadodaria B, Chen X, McGee RB, Hines-Dowell S, Nuccio R, Quinn E, Shurtleff SA, Rusch M, Patel A, Becksfort JB, Wang S, Weaver MS, Ding L, Mardis ER, Wilson RK, Gajjar A, Ellison DW, Pappo AS, Pui CH, Nichols KE, Downing JR. Germline Mutations in Predisposition Genes in Pediatric Cancer. N Engl J Med. 2015 Dec 10;373(24):2336-2346. doi: 10.1056/NEJMoa1508054. Epub 2015 Nov 18. PMID 26580448
- [Background] Mullighan CG, Jeha S, Pei D, Payne-Turner D, Coustan-Smith E, Roberts KG, Waanders E, Choi JK, Ma X, Raimondi SC, Fan Y, Yang W, Song G, Yang JJ, Inaba H, Downing JR, Leung WH, Bowman WP, Relling MV, Evans WE, Zhang J, Campana D, Pui CH. Outcome of children with hypodiploid ALL treated with risk-directed therapy based on MRD levels. Blood. 2015 Dec 24;126(26):2896-9. doi: 10.1182/blood-2015-09-671131. Epub 2015 Nov 2. No abstract available. PMID 26527677
- [Background] Moriyama T, Metzger ML, Wu G, Nishii R, Qian M, Devidas M, Yang W, Cheng C, Cao X, Quinn E, Raimondi S, Gastier-Foster JM, Raetz E, Larsen E, Martin PL, Bowman WP, Winick N, Komada Y, Wang S, Edmonson M, Xu H, Mardis E, Fulton R, Pui CH, Mullighan C, Evans WE, Zhang J, Hunger SP, Relling MV, Nichols KE, Loh ML, Yang JJ. Germline genetic variation in ETV6 and risk of childhood acute lymphoblastic leukaemia: a systematic genetic study. Lancet Oncol. 2015 Dec;16(16):1659-66. doi: 10.1016/S1470-2045(15)00369-1. Epub 2015 Oct 28. PMID 26522332
- [Background] Paugh SW, Coss DR, Bao J, Laudermilk LT, Grace CR, Ferreira AM, Waddell MB, Ridout G, Naeve D, Leuze M, LoCascio PF, Panetta JC, Wilkinson MR, Pui CH, Naeve CW, Uberbacher EC, Bonten EJ, Evans WE. MicroRNAs Form Triplexes with Double Stranded DNA at Sequence-Specific Binding Sites; a Eukaryotic Mechanism via which microRNAs Could Directly Alter Gene Expression. PLoS Comput Biol. 2016 Feb 4;12(2):e1004744. doi: 10.1371/journal.pcbi.1004744. eCollection 2016 Feb. PMID 26844769
- [Background] Iacobucci I, Li Y, Roberts KG, Dobson SM, Kim JC, Payne-Turner D, Harvey RC, Valentine M, McCastlain K, Easton J, Yergeau D, Janke LJ, Shao Y, Chen IM, Rusch M, Zandi S, Kornblau SM, Konopleva M, Jabbour E, Paietta EM, Rowe JM, Pui CH, Gastier-Foster J, Gu Z, Reshmi S, Loh ML, Racevskis J, Tallman MS, Wiernik PH, Litzow MR, Willman CL, McPherson JD, Downing JR, Zhang J, Dick JE, Hunger SP, Mullighan CG. Truncating Erythropoietin Receptor Rearrangements in Acute Lymphoblastic Leukemia. Cancer Cell. 2016 Feb 8;29(2):186-200. doi: 10.1016/j.ccell.2015.12.013. PMID 26859458
- [Background] Hungate EA, Vora SR, Gamazon ER, Moriyama T, Best T, Hulur I, Lee Y, Evans TJ, Ellinghaus E, Stanulla M, Rudant J, Orsi L, Clavel J, Milne E, Scott RJ, Pui CH, Cox NJ, Loh ML, Yang JJ, Skol AD, Onel K. A variant at 9p21.3 functionally implicates CDKN2B in paediatric B-cell precursor acute lymphoblastic leukaemia aetiology. Nat Commun. 2016 Feb 12;7:10635. doi: 10.1038/ncomms10635. PMID 26868379
- [Background] Moriyama T, Nishii R, Perez-Andreu V, Yang W, Klussmann FA, Zhao X, Lin TN, Hoshitsuki K, Nersting J, Kihira K, Hofmann U, Komada Y, Kato M, McCorkle R, Li L, Koh K, Najera CR, Kham SK, Isobe T, Chen Z, Chiew EK, Bhojwani D, Jeffries C, Lu Y, Schwab M, Inaba H, Pui CH, Relling MV, Manabe A, Hori H, Schmiegelow K, Yeoh AE, Evans WE, Yang JJ. NUDT15 polymorphisms alter thiopurine metabolism and hematopoietic toxicity. Nat Genet. 2016 Apr;48(4):367-73. doi: 10.1038/ng.3508. Epub 2016 Feb 15. PMID 26878724
- [Background] Jacola LM, Krull KR, Pui CH, Pei D, Cheng C, Reddick WE, Conklin HM. Longitudinal Assessment of Neurocognitive Outcomes in Survivors of Childhood Acute Lymphoblastic Leukemia Treated on a Contemporary Chemotherapy Protocol. J Clin Oncol. 2016 Apr 10;34(11):1239-47. doi: 10.1200/JCO.2015.64.3205. Epub 2016 Feb 8. PMID 26858334
- [Background] Boland AM, Gibson TM, Lu L, Kaste SC, DeLany JP, Partin RE, Lanctot JQ, Howell CR, Nelson HH, Chemaitilly W, Pui CH, Robison LL, Mulrooney DA, Hudson MM, Ness KK. Dietary Protein Intake and Lean Muscle Mass in Survivors of Childhood Acute Lymphoblastic Leukemia: Report From the St. Jude Lifetime Cohort Study. Phys Ther. 2016 Jul;96(7):1029-38. doi: 10.2522/ptj.20150507. Epub 2016 Feb 18. PMID 26893509
- [Background] Park HW, Tse S, Yang W, Kelly HW, Kaste SC, Pui CH, Relling MV, Tantisira KG. A genetic factor associated with low final bone mineral density in children after a long-term glucocorticoids treatment. Pharmacogenomics J. 2017 Mar;17(2):180-185. doi: 10.1038/tpj.2015.92. Epub 2016 Feb 9. PMID 26856247
- [Background] Vora A, Andreano A, Pui CH, Hunger SP, Schrappe M, Moericke A, Biondi A, Escherich G, Silverman LB, Goulden N, Taskinen M, Pieters R, Horibe K, Devidas M, Locatelli F, Valsecchi MG. Influence of Cranial Radiotherapy on Outcome in Children With Acute Lymphoblastic Leukemia Treated With Contemporary Therapy. J Clin Oncol. 2016 Mar 20;34(9):919-26. doi: 10.1200/JCO.2015.64.2850. Epub 2016 Jan 11. PMID 26755523
- [Background] Wilson CL, Chemaitilly W, Jones KE, Kaste SC, Srivastava DK, Ojha RP, Yasui Y, Pui CH, Robison LL, Hudson MM, Ness KK. Modifiable Factors Associated With Aging Phenotypes Among Adult Survivors of Childhood Acute Lymphoblastic Leukemia. J Clin Oncol. 2016 Jul 20;34(21):2509-15. doi: 10.1200/JCO.2015.64.9525. Epub 2016 Mar 21. PMID 27001572
- [Background] Watts CS, Sciasci JN, Pauley JL, Panetta JC, Pei D, Cheng C, Christensen CM, Mikkelsen TS, Pui CH, Jeha S, Relling MV. Prophylactic Trimethoprim-Sulfamethoxazole Does Not Affect Pharmacokinetics or Pharmacodynamics of Methotrexate. J Pediatr Hematol Oncol. 2016 Aug;38(6):449-52. doi: 10.1097/MPH.0000000000000606. PMID 27322715
- [Background] Liu C, Yang W, Pei D, Cheng C, Smith C, Landier W, Hageman L, Chen Y, Yang JJ, Crews KR, Kornegay N, Karol SE, Wong FL, Jeha S, Sandlund JT, Ribeiro RC, Rubnitz JE, Metzger ML, Pui CH, Evans WE, Bhatia S, Relling MV. Genomewide Approach Validates Thiopurine Methyltransferase Activity Is a Monogenic Pharmacogenomic Trait. Clin Pharmacol Ther. 2017 Mar;101(3):373-381. doi: 10.1002/cpt.463. Epub 2016 Nov 18. PMID 27564568
- [Background] Jacola LM, Edelstein K, Liu W, Pui CH, Hayashi R, Kadan-Lottick NS, Srivastava D, Henderson T, Leisenring W, Robison LL, Armstrong GT, Krull KR. Cognitive, behaviour, and academic functioning in adolescent and young adult survivors of childhood acute lymphoblastic leukaemia: a report from the Childhood Cancer Survivor Study. Lancet Psychiatry. 2016 Oct;3(10):965-972. doi: 10.1016/S2215-0366(16)30283-8. Epub 2016 Sep 14. PMID 27639661
- [Background] Cheung YT, Sabin ND, Reddick WE, Bhojwani D, Liu W, Brinkman TM, Glass JO, Hwang SN, Srivastava D, Pui CH, Robison LL, Hudson MM, Krull KR. Leukoencephalopathy and long-term neurobehavioural, neurocognitive, and brain imaging outcomes in survivors of childhood acute lymphoblastic leukaemia treated with chemotherapy: a longitudinal analysis. Lancet Haematol. 2016 Oct;3(10):e456-e466. doi: 10.1016/S2352-3026(16)30110-7. Epub 2016 Sep 14. PMID 27658980
- [Background] Zhang J, McCastlain K, Yoshihara H, Xu B, Chang Y, Churchman ML, Wu G, Li Y, Wei L, Iacobucci I, Liu Y, Qu C, Wen J, Edmonson M, Payne-Turner D, Kaufmann KB, Takayanagi SI, Wienholds E, Waanders E, Ntziachristos P, Bakogianni S, Wang J, Aifantis I, Roberts KG, Ma J, Song G, Easton J, Mulder HL, Chen X, Newman S, Ma X, Rusch M, Gupta P, Boggs K, Vadodaria B, Dalton J, Liu Y, Valentine ML, Ding L, Lu C, Fulton RS, Fulton L, Tabib Y, Ochoa K, Devidas M, Pei D, Cheng C, Yang J, Evans WE, Relling MV, Pui CH, Jeha S, Harvey RC, Chen IL, Willman CL, Marcucci G, Bloomfield CD, Kohlschmidt J, Mrozek K, Paietta E, Tallman MS, Stock W, Foster MC, Racevskis J, Rowe JM, Luger S, Kornblau SM, Shurtleff SA, Raimondi SC, Mardis ER, Wilson RK, Dick JE, Hunger SP, Loh ML, Downing JR, Mullighan CG; St. Jude Children's Research Hospital-Washington University Pediatric Cancer Genome Project. Deregulation of DUX4 and ERG in acute lymphoblastic leukemia. Nat Genet. 2016 Dec;48(12):1481-1489. doi: 10.1038/ng.3691. Epub 2016 Oct 24. PMID 27776115
- [Background] Pui CH, Pei D, Raimondi SC, Coustan-Smith E, Jeha S, Cheng C, Bowman WP, Sandlund JT, Ribeiro RC, Rubnitz JE, Inaba H, Gruber TA, Leung WH, Yang JJ, Downing JR, Evans WE, Relling MV, Campana D. Clinical impact of minimal residual disease in children with different subtypes of acute lymphoblastic leukemia treated with Response-Adapted therapy. Leukemia. 2017 Feb;31(2):333-339. doi: 10.1038/leu.2016.234. Epub 2016 Aug 18. PMID 27560110
- [Background] Qian M, Zhang H, Kham SK, Liu S, Jiang C, Zhao X, Lu Y, Goodings C, Lin TN, Zhang R, Moriyama T, Yin Z, Li Z, Quah TC, Ariffin H, Tan AM, Shen S, Bhojwani D, Hu S, Chen S, Zheng H, Pui CH, Yeoh AE, Yang JJ. Whole-transcriptome sequencing identifies a distinct subtype of acute lymphoblastic leukemia with predominant genomic abnormalities of EP300 and CREBBP. Genome Res. 2017 Feb;27(2):185-195. doi: 10.1101/gr.209163.116. Epub 2016 Nov 30. PMID 27903646
- [Background] Cheung YT, Chemaitilly W, Mulrooney DA, Brinkman TM, Liu W, Banerjee P, Srivastava D, Pui CH, Robison LL, Hudson MM, Krull KR. Association between dehydroepiandrosterone-sulfate and attention in long-term survivors of childhood acute lymphoblastic leukemia treated with only chemotherapy. Psychoneuroendocrinology. 2017 Feb;76:114-118. doi: 10.1016/j.psyneuen.2016.11.014. Epub 2016 Nov 16. PMID 27907849
- [Background] Inaba H, Pei D, Wolf J, Howard SC, Hayden RT, Go M, Varechtchouk O, Hahn T, Buaboonnam J, Metzger ML, Rubnitz JE, Ribeiro RC, Sandlund JT, Jeha S, Cheng C, Evans WE, Relling MV, Pui CH. Infection-related complications during treatment for childhood acute lymphoblastic leukemia. Ann Oncol. 2017 Feb 1;28(2):386-392. doi: 10.1093/annonc/mdw557. PMID 28426102
- [Background] Eissa HM, Zhou Y, Panetta JC, Browne EK, Jeha S, Cheng C, Relling MV, Campana D, Pui CH, Inaba H. The effect of body mass index at diagnosis on clinical outcome in children with newly diagnosed acute lymphoblastic leukemia. Blood Cancer J. 2017 Feb 17;7(2):e531. doi: 10.1038/bcj.2017.11. PMID 28212374
- [Background] Portera MV, Karol SE, Smith C, Yang W, Cheng C, Neel MD, Pui CH, Relling MV, Kaste SC. Osteonecrosis is unrelated to hip anatomy in children with acute lymphoblastic leukemia. Pediatr Blood Cancer. 2017 Jul;64(7):10.1002/pbc.26407. doi: 10.1002/pbc.26407. Epub 2016 Dec 30. PMID 28035753
- [Background] Liu Y, Fernandez CA, Smith C, Yang W, Cheng C, Panetta JC, Kornegay N, Liu C, Ramsey LB, Karol SE, Janke LJ, Larsen EC, Winick N, Carroll WL, Loh ML, Raetz EA, Hunger SP, Devidas M, Yang JJ, Mullighan CG, Zhang J, Evans WE, Jeha S, Pui CH, Relling MV. Genome-Wide Study Links PNPLA3 Variant With Elevated Hepatic Transaminase After Acute Lymphoblastic Leukemia Therapy. Clin Pharmacol Ther. 2017 Jul;102(1):131-140. doi: 10.1002/cpt.629. Epub 2017 Apr 4. PMID 28090653
- [Background] Karol SE, Larsen E, Cheng C, Cao X, Yang W, Ramsey LB, Fernandez CA, McCorkle JR, Paugh SW, Autry RJ, Lopez-Lopez E, Diouf B, Jeha S, Pui CH, Raetz EA, Winick NJ, Carroll WL, Hunger SP, Loh ML, Devidas M, Evans WE, Yang JJ, Relling MV. Genetics of ancestry-specific risk for relapse in acute lymphoblastic leukemia. Leukemia. 2017 Jun;31(6):1325-1332. doi: 10.1038/leu.2017.24. Epub 2017 Jan 18. PMID 28096535
- [Background] Nassar SL, Conklin HM, Zhou Y, Ashford JM, Reddick WE, Glass JO, Laningham FH, Jeha S, Cheng C, Pui CH. Neurocognitive outcomes among children who experienced seizures during treatment for acute lymphoblastic leukemia. Pediatr Blood Cancer. 2017 Aug;64(8):10.1002/pbc.26436. doi: 10.1002/pbc.26436. Epub 2017 Jan 28. PMID 28130818
- [Background] Cheung YT, Brinkman TM, Mulrooney DA, Mzayek Y, Liu W, Banerjee P, Panoskaltsis-Mortari A, Srivastava D, Pui CH, Robison LL, Hudson MM, Krull KR. Impact of sleep, fatigue, and systemic inflammation on neurocognitive and behavioral outcomes in long-term survivors of childhood acute lymphoblastic leukemia. Cancer. 2017 Sep 1;123(17):3410-3419. doi: 10.1002/cncr.30742. Epub 2017 Apr 27. PMID 28452142
- [Background] Hu S, Qian M, Zhang H, Guo Y, Yang J, Zhao X, He H, Lu J, Pan J, Chang M, Du G, Lin TN, Kham SK, Quah TC, Ariffin H, Tan AM, Cheng Y, Li C, Yeoh AE, Pui CH, Skanderup AJ, Yang JJ. Whole-genome noncoding sequence analysis in T-cell acute lymphoblastic leukemia identifies oncogene enhancer mutations. Blood. 2017 Jun 15;129(24):3264-3268. doi: 10.1182/blood-2017-03-771162. Epub 2017 Apr 13. PMID 28408461
- [Background] Karol SE, Yang W, Smith C, Cheng C, Stewart CF, Baker SD, Sandlund JT, Rubnitz JE, Bishop MW, Pappo AS, Jeha S, Pui CH, Relling MV. Palmar-plantar erythrodysesthesia syndrome following treatment with high-dose methotrexate or high-dose cytarabine. Cancer. 2017 Sep 15;123(18):3602-3608. doi: 10.1002/cncr.30762. Epub 2017 May 11. PMID 28493546
- [Background] Ramsey LB, Pounds S, Cheng C, Cao X, Yang W, Smith C, Karol SE, Liu C, Panetta JC, Inaba H, Rubnitz JE, Metzger ML, Ribeiro RC, Sandlund JT, Jeha S, Pui CH, Evans WE, Relling MV. Genetics of pleiotropic effects of dexamethasone. Pharmacogenet Genomics. 2017 Aug;27(8):294-302. doi: 10.1097/FPC.0000000000000293. PMID 28628558
- [Background] Moriyama T, Yang YL, Nishii R, Ariffin H, Liu C, Lin TN, Yang W, Lin DT, Yu CH, Kham S, Pui CH, Evans WE, Jeha S, Relling MV, Yeoh AE, Yang JJ. Novel variants in NUDT15 and thiopurine intolerance in children with acute lymphoblastic leukemia from diverse ancestry. Blood. 2017 Sep 7;130(10):1209-1212. doi: 10.1182/blood-2017-05-782383. Epub 2017 Jun 28. PMID 28659275
- [Background] Green DM, Zhu L, Wang M, Chemaitilly W, Srivastava D, Kutteh WH, Ke RW, Sklar CA, Pui CH, Kun LE, Ribeiro RC, Robison LL, Hudson MM. Effect of cranial irradiation on sperm concentration of adult survivors of childhood acute lymphoblastic leukemia: a report from the St. Jude Lifetime Cohort Studydagger. Hum Reprod. 2017 Jun 1;32(6):1192-1201. doi: 10.1093/humrep/dex082. PMID 28444255
- [Background] Chemaitilly W, Li Z, Krasin MJ, Brooke RJ, Wilson CL, Green DM, Klosky JL, Barnes N, Clark KL, Farr JB, Fernandez-Pineda I, Bishop MW, Metzger M, Pui CH, Kaste SC, Ness KK, Srivastava DK, Robison LL, Hudson MM, Yasui Y, Sklar CA. Premature Ovarian Insufficiency in Childhood Cancer Survivors: A Report From the St. Jude Lifetime Cohort. J Clin Endocrinol Metab. 2017 Jul 1;102(7):2242-2250. doi: 10.1210/jc.2016-3723. PMID 28368472
- [Background] Bainer RO, Trendowski MR, Cheng C, Pei D, Yang W, Paugh SW, Goss KH, Skol AD, Pavlidis P, Pui CH, Gilliam TC, Evans WE, Onel K. A p53-regulated apoptotic gene signature predicts treatment response and outcome in pediatric acute lymphoblastic leukemia. Cancer Manag Res. 2017 Sep 13;9:397-410. doi: 10.2147/CMAR.S139864. eCollection 2017. PMID 28979163
- [Background] Wolf J, Tang L, Flynn PM, Pui CH, Gaur AH, Sun Y, Inaba H, Stewart T, Hayden RT, Hakim H, Jeha S. Levofloxacin Prophylaxis During Induction Therapy for Pediatric Acute Lymphoblastic Leukemia. Clin Infect Dis. 2017 Nov 13;65(11):1790-1798. doi: 10.1093/cid/cix644. PMID 29020310
- [Background] Qian M, Cao X, Devidas M, Yang W, Cheng C, Dai Y, Carroll A, Heerema NA, Zhang H, Moriyama T, Gastier-Foster JM, Xu H, Raetz E, Larsen E, Winick N, Bowman WP, Martin PL, Mardis ER, Fulton R, Zambetti G, Borowitz M, Wood B, Nichols KE, Carroll WL, Pui CH, Mullighan CG, Evans WE, Hunger SP, Relling MV, Loh ML, Yang JJ. TP53 Germline Variations Influence the Predisposition and Prognosis of B-Cell Acute Lymphoblastic Leukemia in Children. J Clin Oncol. 2018 Feb 20;36(6):591-599. doi: 10.1200/JCO.2017.75.5215. Epub 2018 Jan 4. PMID 29300620
- [Background] Howell CR, Wilson CL, Ehrhardt MJ, Partin RE, Kaste SC, Lanctot JQ, Pui CH, Robison LL, Hudson MM, Ness KK. Clinical impact of sedentary behaviors in adult survivors of acute lymphoblastic leukemia: A report from the St. Jude Lifetime Cohort study. Cancer. 2018 Mar 1;124(5):1036-1043. doi: 10.1002/cncr.31162. Epub 2017 Dec 4. PMID 29205290
- [Background] Inaba H, Cao X, Han AQ, Panetta JC, Ness KK, Metzger ML, Rubnitz JE, Ribeiro RC, Sandlund JT, Jeha S, Cheng C, Pui CH, Relling MV, Kaste SC. Bone mineral density in children with acute lymphoblastic leukemia. Cancer. 2018 Mar 1;124(5):1025-1035. doi: 10.1002/cncr.31184. Epub 2017 Dec 19. PMID 29266176
- [Background] Churchman ML, Qian M, Te Kronnie G, Zhang R, Yang W, Zhang H, Lana T, Tedrick P, Baskin R, Verbist K, Peters JL, Devidas M, Larsen E, Moore IM, Gu Z, Qu C, Yoshihara H, Porter SN, Pruett-Miller SM, Wu G, Raetz E, Martin PL, Bowman WP, Winick N, Mardis E, Fulton R, Stanulla M, Evans WE, Relling MV, Pui CH, Hunger SP, Loh ML, Handgretinger R, Nichols KE, Yang JJ, Mullighan CG. Germline Genetic IKZF1 Variation and Predisposition to Childhood Acute Lymphoblastic Leukemia. Cancer Cell. 2018 May 14;33(5):937-948.e8. doi: 10.1016/j.ccell.2018.03.021. Epub 2018 Apr 19. PMID 29681510
- [Background] Zhang Y, Gao Y, Zhang H, Zhang J, He F, Hnizda A, Qian M, Liu X, Gocho Y, Pui CH, Cheng T, Wang Q, Yang JJ, Zhu X, Liu X. PDGFRB mutation and tyrosine kinase inhibitor resistance in Ph-like acute lymphoblastic leukemia. Blood. 2018 May 17;131(20):2256-2261. doi: 10.1182/blood-2017-11-817510. Epub 2018 Feb 6. PMID 29434033
- [Background] Pui CH, Yang JJ, Bhakta N, Rodriguez-Galindo C. Global efforts toward the cure of childhood acute lymphoblastic leukaemia. Lancet Child Adolesc Health. 2018 Jun;2(6):440-454. doi: 10.1016/S2352-4642(18)30066-X. Epub 2018 Mar 30. PMID 30169285
- [Background] Liu W, Cheung YT, Conklin HM, Jacola LM, Srivastava D, Nolan VG, Zhang H, Gurney JG, Huang IC, Robison LL, Pui CH, Hudson MM, Krull KR. Evolution of neurocognitive function in long-term survivors of childhood acute lymphoblastic leukemia treated with chemotherapy only. J Cancer Surviv. 2018 Jun;12(3):398-406. doi: 10.1007/s11764-018-0679-7. Epub 2018 Feb 27. PMID 29484542
- [Background] Liu W, Cheung YT, Brinkman TM, Banerjee P, Srivastava D, Nolan VG, Zhang H, Gurney JG, Pui CH, Robison LL, Hudson MM, Krull KR. Behavioral symptoms and psychiatric disorders in child and adolescent long-term survivors of childhood acute lymphoblastic leukemia treated with chemotherapy only. Psychooncology. 2018 Jun;27(6):1597-1607. doi: 10.1002/pon.4699. Epub 2018 Mar 30. PMID 29521470
- [Background] Cheung YT, Khan RB, Liu W, Brinkman TM, Edelmann MN, Reddick WE, Pei D, Panoskaltsis-Mortari A, Srivastava D, Cheng C, Robison LL, Hudson MM, Pui CH, Krull KR. Association of Cerebrospinal Fluid Biomarkers of Central Nervous System Injury With Neurocognitive and Brain Imaging Outcomes in Children Receiving Chemotherapy for Acute Lymphoblastic Leukemia. JAMA Oncol. 2018 Jul 12;4(7):e180089. doi: 10.1001/jamaoncol.2018.0089. Epub 2018 Jul 12. PMID 29596541
- [Background] Hakim H, Dallas R, Wolf J, Tang L, Schultz-Cherry S, Darling V, Johnson C, Karlsson EA, Chang TC, Jeha S, Pui CH, Sun Y, Pounds S, Hayden RT, Tuomanen E, Rosch JW. Gut Microbiome Composition Predicts Infection Risk During Chemotherapy in Children With Acute Lymphoblastic Leukemia. Clin Infect Dis. 2018 Aug 1;67(4):541-548. doi: 10.1093/cid/ciy153. PMID 29518185
- [Background] Varedi M, Lu L, Howell CR, Partin RE, Hudson MM, Pui CH, Krull KR, Robison LL, Ness KK, McKenna RF. Peripheral Neuropathy, Sensory Processing, and Balance in Survivors of Acute Lymphoblastic Leukemia. J Clin Oncol. 2018 Aug 1;36(22):2315-2322. doi: 10.1200/JCO.2017.76.7871. Epub 2018 May 29. PMID 29812998
- [Background] Huang IC, Brinkman TM, Mullins L, Pui CH, Robison LL, Hudson MM, Krull KR. Child symptoms, parent behaviors, and family strain in long-term survivors of childhood acute lymphoblastic leukemia. Psychooncology. 2018 Aug;27(8):2031-2038. doi: 10.1002/pon.4769. Epub 2018 Jun 29. PMID 29772082
- [Background] Kesler SR, Ogg R, Reddick WE, Phillips N, Scoggins M, Glass JO, Cheung YT, Pui CH, Robison LL, Hudson MM, Krull KR. Brain Network Connectivity and Executive Function in Long-Term Survivors of Childhood Acute Lymphoblastic Leukemia. Brain Connect. 2018 Aug;8(6):333-342. doi: 10.1089/brain.2017.0574. PMID 29936880
- [Background] Alexander TB, Gu Z, Iacobucci I, Dickerson K, Choi JK, Xu B, Payne-Turner D, Yoshihara H, Loh ML, Horan J, Buldini B, Basso G, Elitzur S, de Haas V, Zwaan CM, Yeoh A, Reinhardt D, Tomizawa D, Kiyokawa N, Lammens T, De Moerloose B, Catchpoole D, Hori H, Moorman A, Moore AS, Hrusak O, Meshinchi S, Orgel E, Devidas M, Borowitz M, Wood B, Heerema NA, Carrol A, Yang YL, Smith MA, Davidsen TM, Hermida LC, Gesuwan P, Marra MA, Ma Y, Mungall AJ, Moore RA, Jones SJM, Valentine M, Janke LJ, Rubnitz JE, Pui CH, Ding L, Liu Y, Zhang J, Nichols KE, Downing JR, Cao X, Shi L, Pounds S, Newman S, Pei D, Guidry Auvil JM, Gerhard DS, Hunger SP, Inaba H, Mullighan CG. The genetic basis and cell of origin of mixed phenotype acute leukaemia. Nature. 2018 Oct;562(7727):373-379. doi: 10.1038/s41586-018-0436-0. Epub 2018 Sep 12. PMID 30209392
- [Background] Sabin ND, Cheung YT, Reddick WE, Bhojwani D, Liu W, Glass JO, Brinkman TM, Hwang SN, Srivastava D, Pui CH, Robison LL, Hudson MM, Krull KR. The Impact of Persistent Leukoencephalopathy on Brain White Matter Microstructure in Long-Term Survivors of Acute Lymphoblastic Leukemia Treated with Chemotherapy Only. AJNR Am J Neuroradiol. 2018 Oct;39(10):1919-1925. doi: 10.3174/ajnr.A5791. Epub 2018 Sep 13. PMID 30213807
- [Background] Cheung YT, Eskind A, Inaba H, Hudson MM, Pui CH, Krull KR, Wolf J. Association of Bacteremic Sepsis With Long-term Neurocognitive Dysfunction in Pediatric Patients With Acute Lymphoblastic Leukemia. JAMA Pediatr. 2018 Nov 1;172(11):1092-1095. doi: 10.1001/jamapediatrics.2018.2500. PMID 30264151
- [Background] Browne EK, Zhou Y, Chemaitilly W, Panetta JC, Ness KK, Kaste SC, Cheng C, Relling MV, Pui CH, Inaba H. Changes in body mass index, height, and weight in children during and after therapy for acute lymphoblastic leukemia. Cancer. 2018 Nov 1;124(21):4248-4259. doi: 10.1002/cncr.31736. Epub 2018 Oct 25. PMID 30358906
- [Background] Wilson CL, Howell CR, Partin RE, Lu L, Kaste SC, Mulrooney DA, Pui CH, Lanctot JQ, Srivastava DK, Robison LL, Hudson MM, Ness KK. Influence of fitness on health status among survivors of acute lymphoblastic leukemia. Pediatr Blood Cancer. 2018 Nov;65(11):e27286. doi: 10.1002/pbc.27286. Epub 2018 Jul 29. PMID 30058279
- [Background] Li JF, Dai YT, Lilljebjorn H, Shen SH, Cui BW, Bai L, Liu YF, Qian MX, Kubota Y, Kiyoi H, Matsumura I, Miyazaki Y, Olsson L, Tan AM, Ariffin H, Chen J, Takita J, Yasuda T, Mano H, Johansson B, Yang JJ, Yeoh AE, Hayakawa F, Chen Z, Pui CH, Fioretos T, Chen SJ, Huang JY. Transcriptional landscape of B cell precursor acute lymphoblastic leukemia based on an international study of 1,223 cases. Proc Natl Acad Sci U S A. 2018 Dec 11;115(50):E11711-E11720. doi: 10.1073/pnas.1814397115. Epub 2018 Nov 28. PMID 30487223
- [Background] Green DM, Wang M, Krasin MJ, Srivastava D, Relling MV, Howell CR, Ness KK, Kaste SC, Greene W, Jay DW, Fernandez-Pineda I, Pui CH, Jeha S, Bishop MW, Furman WL, Robison LL, Hudson MM. Serum Alanine Aminotransferase Elevations in Survivors of Childhood Cancer: A Report From the St. Jude Lifetime Cohort Study. Hepatology. 2019 Jan;69(1):94-106. doi: 10.1002/hep.30176. Epub 2018 Dec 25. PMID 30016547
- [Background] Fellah S, Cheung YT, Scoggins MA, Zou P, Sabin ND, Pui CH, Robison LL, Hudson MM, Ogg RJ, Krull KR. Brain Activity Associated With Attention Deficits Following Chemotherapy for Childhood Acute Lymphoblastic Leukemia. J Natl Cancer Inst. 2019 Feb 1;111(2):201-209. doi: 10.1093/jnci/djy089. PMID 29790971
- [Background] Qian M, Xu H, Perez-Andreu V, Roberts KG, Zhang H, Yang W, Zhang S, Zhao X, Smith C, Devidas M, Gastier-Foster JM, Raetz E, Larsen E, Burchard EG, Winick N, Bowman WP, Martin PL, Borowitz M, Wood B, Antillon-Klussmann F, Pui CH, Mullighan CG, Evans WE, Hunger SP, Relling MV, Loh ML, Yang JJ. Novel susceptibility variants at the ERG locus for childhood acute lymphoblastic leukemia in Hispanics. Blood. 2019 Feb 14;133(7):724-729. doi: 10.1182/blood-2018-07-862946. Epub 2018 Dec 3. PMID 30510082
- [Background] Gu Z, Churchman ML, Roberts KG, Moore I, Zhou X, Nakitandwe J, Hagiwara K, Pelletier S, Gingras S, Berns H, Payne-Turner D, Hill A, Iacobucci I, Shi L, Pounds S, Cheng C, Pei D, Qu C, Newman S, Devidas M, Dai Y, Reshmi SC, Gastier-Foster J, Raetz EA, Borowitz MJ, Wood BL, Carroll WL, Zweidler-McKay PA, Rabin KR, Mattano LA, Maloney KW, Rambaldi A, Spinelli O, Radich JP, Minden MD, Rowe JM, Luger S, Litzow MR, Tallman MS, Racevskis J, Zhang Y, Bhatia R, Kohlschmidt J, Mrozek K, Bloomfield CD, Stock W, Kornblau S, Kantarjian HM, Konopleva M, Evans WE, Jeha S, Pui CH, Yang J, Paietta E, Downing JR, Relling MV, Zhang J, Loh ML, Hunger SP, Mullighan CG. PAX5-driven subtypes of B-progenitor acute lymphoblastic leukemia. Nat Genet. 2019 Feb;51(2):296-307. doi: 10.1038/s41588-018-0315-5. Epub 2019 Jan 14. PMID 30643249
- [Background] Teachey DT, Pui CH. Comparative features and outcomes between paediatric T-cell and B-cell acute lymphoblastic leukaemia. Lancet Oncol. 2019 Mar;20(3):e142-e154. doi: 10.1016/S1470-2045(19)30031-2. PMID 30842058
- [Background] Pui CH, Rebora P, Schrappe M, Attarbaschi A, Baruchel A, Basso G, Cave H, Elitzur S, Koh K, Liu HC, Paulsson K, Pieters R, Silverman LB, Stary J, Vora A, Yeoh A, Harrison CJ, Valsecchi MG; Ponte di Legno Childhood ALL Working Group. Outcome of Children With Hypodiploid Acute Lymphoblastic Leukemia: A Retrospective Multinational Study. J Clin Oncol. 2019 Apr 1;37(10):770-779. doi: 10.1200/JCO.18.00822. Epub 2019 Jan 18. PMID 30657737
- [Background] Qian M, Zhao X, Devidas M, Yang W, Gocho Y, Smith C, Gastier-Foster JM, Li Y, Xu H, Zhang S, Jeha S, Zhai X, Sanda T, Winter SS, Dunsmore KP, Raetz EA, Carroll WL, Winick NJ, Rabin KR, Zweidler-Mckay PA, Wood B, Pui CH, Evans WE, Hunger SP, Mullighan CG, Relling MV, Loh ML, Yang JJ. Genome-Wide Association Study of Susceptibility Loci for T-Cell Acute Lymphoblastic Leukemia in Children. J Natl Cancer Inst. 2019 Dec 1;111(12):1350-1357. doi: 10.1093/jnci/djz043. PMID 30938820
- [Background] Pui CH, Nichols KE, Yang JJ. Somatic and germline genomics in paediatric acute lymphoblastic leukaemia. Nat Rev Clin Oncol. 2019 Apr;16(4):227-240. doi: 10.1038/s41571-018-0136-6. PMID 30546053
- [Background] Krull KR, Li C, Phillips NS, Cheung YT, Brinkman TM, Wilson CL, Armstrong GT, Khan RB, Merchant TE, Sabin ND, Srivastava D, Pui CH, Robison LL, Hudson MM, Sklar CA, Chemaitilly W. Growth hormone deficiency and neurocognitive function in adult survivors of childhood acute lymphoblastic leukemia. Cancer. 2019 May 15;125(10):1748-1755. doi: 10.1002/cncr.31975. Epub 2019 Jan 28. PMID 30690723
- [Background] Mulrooney DA, Hyun G, Ness KK, Bhakta N, Pui CH, Ehrhardt MJ, Krull KR, Crom DB, Chemaitilly W, Srivastava DK, Relling MV, Jeha S, Green DM, Yasui Y, Robison LL, Hudson MM. The changing burden of long-term health outcomes in survivors of childhood acute lymphoblastic leukaemia: a retrospective analysis of the St Jude Lifetime Cohort Study. Lancet Haematol. 2019 Jun;6(6):e306-e316. doi: 10.1016/S2352-3026(19)30050-X. Epub 2019 May 8. PMID 31078468
- [Background] Robinson KM, Yang W, Karol SE, Kornegay N, Jay D, Cheng C, Choi JK, Campana D, Pui CH, Wood B, Borowitz MJ, Gastier-Foster J, Larsen EC, Winick N, Carroll WL, Loh ML, Raetz EA, Hunger SP, Devidas M, Mardis ER, Fulton RS, Relling MV, Jeha S. No evidence that G6PD deficiency affects the efficacy or safety of daunorubicin in acute lymphoblastic leukemia induction therapy. Pediatr Blood Cancer. 2019 Jun;66(6):e27681. doi: 10.1002/pbc.27681. Epub 2019 Mar 7. PMID 30848065
- [Background] Finch ER, Janke LJ, Smith CA, Karol SE, Pei D, Cheng C, Kaste SC, Inaba H, Pui CH, Wolf J, Relling MV. Bloodstream infections exacerbate incidence and severity of symptomatic glucocorticoid-induced osteonecrosis. Pediatr Blood Cancer. 2019 Jun;66(6):e27669. doi: 10.1002/pbc.27669. Epub 2019 Feb 13. PMID 30758124
- [Background] Sharkey CM, Clawson AH, Mullins LL, Brinkman TM, Pui CH, Hudson MM, Krull KR. The relationship of child executive functions to parenting capacities in childhood acute lymphoblastic leukemia survivors. Pediatr Blood Cancer. 2019 Aug;66(8):e27761. doi: 10.1002/pbc.27761. Epub 2019 Apr 29. PMID 31033172
- [Derived] Purvis K, Zhou Y, Karol SE, Rubnitz JE, Ribeiro RC, Lee S, Yang JJ, Bowman WP, Wang L, Dixon SB, Roberts KG, Gao Q, Cheng C, Mullighan CG, Jeha S, Pui CH, Inaba H. Outcomes in patients with ETV6::RUNX1 or high-hyperdiploid B-ALL treated in the St. Jude Total Therapy XV/XVI studies. Blood. 2025 Jan 9;145(2):190-201. doi: 10.1182/blood.2024024936. PMID 39316653
- [Derived] Chang TC, Chen W, Qu C, Cheng Z, Hedges D, Elsayed A, Pounds SB, Shago M, Rabin KR, Raetz EA, Devidas M, Cheng C, Angiolillo A, Baviskar P, Borowitz M, Burke MJ, Carroll A, Carroll WL, Chen IM, Harvey R, Heerema N, Iacobucci I, Wang JR, Jeha S, Larsen E, Mattano L, Maloney K, Pui CH, Ramirez NC, Salzer W, Willman C, Winick N, Wood B, Hunger SP, Wu G, Mullighan CG, Loh ML. Genomic Determinants of Outcome in Acute Lymphoblastic Leukemia. J Clin Oncol. 2024 Oct 10;42(29):3491-3503. doi: 10.1200/JCO.23.02238. Epub 2024 Aug 9. PMID 39121442
- [Derived] Escherich CS, Chen W, Li Y, Yang W, Nishii R, Li Z, Raetz EA, Devidas M, Wu G, Nichols KE, Inaba H, Pui CH, Jeha S, Camitta BM, Larsen E, Hunger SP, Loh ML, Yang JJ. Germ line genetic NBN variation and predisposition to B-cell acute lymphoblastic leukemia in children. Blood. 2024 May 30;143(22):2270-2283. doi: 10.1182/blood.2023023336. PMID 38446568
- [Derived] Partanen M, Alberts NM, Conklin HM, Krull KR, Pui CH, Anghelescu DA, Jacola LM. Neuropathic pain and neurocognitive functioning in children treated for acute lymphoblastic leukemia. Pain. 2022 Jun 1;163(6):1070-1077. doi: 10.1097/j.pain.0000000000002485. Epub 2021 Sep 25. PMID 34813516
- [Derived] Finch ER, Smith CA, Yang W, Liu Y, Kornegay NM, Panetta JC, Crews KR, Molinelli AR, Cheng C, Pei D, Ramsey LB, Karol SE, Inaba H, Sandlund JT, Metzger M, Evans WE, Jeha S, Pui CH, Relling MV. Asparaginase formulation impacts hypertriglyceridemia during therapy for acute lymphoblastic leukemia. Pediatr Blood Cancer. 2020 Jan;67(1):e28040. doi: 10.1002/pbc.28040. Epub 2019 Oct 14. PMID 31612640
- [Derived] Liu Y, Smith CA, Panetta JC, Yang W, Thompson LE, Counts JP, Molinelli AR, Pei D, Kornegay NM, Crews KR, Swanson H, Cheng C, Karol SE, Evans WE, Inaba H, Pui CH, Jeha S, Relling MV. Antibodies Predict Pegaspargase Allergic Reactions and Failure of Rechallenge. J Clin Oncol. 2019 Aug 10;37(23):2051-2061. doi: 10.1200/JCO.18.02439. Epub 2019 Jun 12. PMID 31188727
- [Derived] Faham M, Zheng J, Moorhead M, Carlton VE, Stow P, Coustan-Smith E, Pui CH, Campana D. Deep-sequencing approach for minimal residual disease detection in acute lymphoblastic leukemia. Blood. 2012 Dec 20;120(26):5173-80. doi: 10.1182/blood-2012-07-444042. Epub 2012 Oct 16. PMID 23074282
- See also: St Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 501 patients were recruited between June 2000 and October 2007.
Pre-assignment Details: 501 patients were enrolled on the study. 3 patients were determined to be ineligible shortly after enrollment (wrong diagnosis - AML or CML in blast crisis).498 patients started the study.
Groups:
- Total Therapy: Total therapy applies to all eligible patients and includes remission induction, consolidation, and continuation therapy.
- 4 hr: 4 hour High-Dose Methotrexate Infusion in upfront window treatment
- 24 hr: 24 hour High-Dose Methotrexate Infusion in upfront window treatment
- Non Randomized: Patients not randomized for window study
Period: Window Therapy
Arm/Group | Total Therapy | 4 hr | 24 hr | Non Randomized
Started | 0 | 176 | 180 | 142
Completed | 0 | 176 | 180 | 142
Not Completed | 0 | 0 | 0 | 0
Period: Total Therapy
Arm/Group | Total Therapy | 4 hr | 24 hr | Non Randomized
Started | 498 | 0 | 0 | 0
Completed | 458 | 0 | 0 | 0
Not Completed | 40 | 0 | 0 | 0
Not completed — Death | 35 | 0 | 0 | 0
Not completed — Non Compliance | 5 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Total Therapy | 4 hr | 24 hr | Non Randomized | Total
Number analyzed (Participants) | 498 | 0 | 0 | 0 | 498
Age, Customized [Number; unit: participants] — Prior experience indicate different responses for children under the age of ten and those who are 10 and older.
  participants
    1 to 9 years | 372 |  |  |  | 372
    >=10 years | 126 |  |  |  | 126
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 219 |  |  |  | 219
  Male | 279 |  |  |  | 279

OUTCOME MEASURES:

1. Primary Outcome: Overall Event-free Survival (EFS)
Description: EFS was measured from the start of on-study to the date of first treatment failure of any kind (relapse, death, lineage switch, or second malignancy) or to the last date of follow-up. Failure to enter remission was considered an event at time zero. Measurement was determined by Kaplan-Meyer estimate.
Time Frame: Median follow-up time (range) 5.6 (1.3 to 8.9) years
Population: 498 enrolled patients were eligible for analysis to estimate the overall event-free survival of children at least one year of age at diagnosis who are treated with risk-directed therapy.
Measure: Number; unit: Percentage of Participants
Groups:
- Total Therapy: Total therapy applies to all eligible patients.
Arm/Group | Total Therapy
Number analyzed (Participants) | 498
Percentage of Participants | 87.3 [.831 to .901]

2. Primary Outcome: Continuous Complete Remission Since Week 56 Therapy.
Description: CCR was measured from end of week 56 therapy to the date of first treatment failure of any kind (relapse, death, lineage switch, or second malignancy) or to the last date of follow-up. Measurement was determined by Kaplan-Meyer estimate.
Time Frame: Median follow up time (range) 4.5 (1 to 7.8) years
Population: Patients meeting the following high risk CNS Relapse criteria: white cell blood cell count at diagnosis more than 100,000; Philadelphia Chromosome Positive; CNS 3 at diagnosis; T-Lineage with white blood cell count more than 50,000.
Measure: Number; unit: Percentage of participants
Groups:
- Patients With High Risk of CNS Relapse: This is a subset of all patients enrolled. It is not a specific treatment arm.
Arm/Group | Patients With High Risk of CNS Relapse
Number analyzed (Participants) | 70
Percentage of participants | 92.2 [82 to 100]

3. Secondary Outcome: Minimal Residual Disease (MRD)
Description: Detection of MRD at end of induction where positive MRD was defined as one or more leukemic cell per 10,000 mononuclear bone-marrow cells (>=0.01%).
Time Frame: End of Induction (Day 46 MRD measurement)
Population: Patients who completed induction and had successful MRD studies on day 46.
Measure: Number; unit: participants
Arm/Group | Total Therapy
Number analyzed (Participants) | 492
participants
  Negative <0.01% | 390
  Positive >= 0.01% | 102
Statistical Analysis 1: Comparison: Total Therapy; Of the 498 eligible patients, 492 were successfully evaluated with day 46 MRD measurement; Test type: Superiority or Other; Binomial proportion; Binomial proportion = 79.27, 95% CI 2-sided [75.69 to 82.85]

4. Secondary Outcome: Mean Difference of Active Methotrexate Polyglutamates (MTXPG) in Leukemia Cells Between Two Arms (4 Hours vs. 24 Hours).
Description: Children were randomly assigned to receive initial single-agent treatment with HDMTX (1g/m^2) as either a 24-hour infusion or a 4-hour infusion and the outcome measure was the accumulation of MTXPG in leukemia cells.
Time Frame: 42 hours after start of high dose methotrexate infusion (HDMTX)
Population: The 286 patients randomized to treatment with high-dose methotrexate (HDMTX) who had methotrexate polyglutamate (MTXPG) concentration measured in bone marrow ALL cells .
Measure: Mean (Standard Deviation); unit: pmol/1,000,000,000 cells
Arm/Group | 4 hr | 24 hr
Number analyzed (Participants) | 136 | 150
pmol/1,000,000,000 cells | 1688 (2015) | 2521 (2950)
Statistical Analysis 1: Comparison: 4 hr vs 24 hr; t-test stratified for lineage and ploidy; Test type: Superiority or Other; p = .0062, t-test, 2 sided — p-value from t-test after stratified for lineage and ploidy

5. Secondary Outcome: Circulating Leukemia Cells in Peripheral Blood Change From Prior to the Methotrexate Infusion to Three Days After Between Two Arms (4 Hours vs. 24 Hours)
Description: White blood cell (leukocytes) counts in peripheral blood by Complete Blood Count
  Measurement: Percentage change of leukemia cells from baseline
Time Frame: Immediately before the methotrexate infusion and three days after subsequent infusion
Population: Three hundred twenty (320) patients were evaluable to assess the influence of infusion duration on methotrexate's antileukemic effects.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | 4 hr | 24 hr
Number analyzed (Participants) | 156 | 164
Percent change | -44 (42.2) | -50 (35.5)
Statistical Analysis 1: Comparison: 4 hr vs 24 hr; t-test adjusting for lineage and ploidy; Test type: Superiority or Other; p = .15, t-test, 2 sided — p-value from t-test after adjusted for lineage and ploidy

6. Other Pre Specified Outcome: Median Difference in CASP1 Gene Expression in Primary Leukemia Cells of Patients in Glucocorticoid-resistant Cells vs Glucocorticoid-sensitive Cells
Description: Prednisolone sensitivity was measured in primary leukemia cells from bone marrow collected at diagnosis. Expression of CASP1 was determined by HG-U133A microarray. Values given are gene expression values, and the unit is arbitrary units (AU) defined as scaled fluorescence measured on microarray.
Time Frame: Pre-treatment
Population: One hundred forty-four (144) patients were evaluable to assess prednisolone sensitivity measured in bone marrow ALL cells and CASP1 expression in RNA by MTT assay.
Measure: Median (Inter-Quartile Range); unit: arbitrary units
Arm/Group | Total Therapy
Number analyzed (Participants) | 144
arbitrary units
  Prednisolone-sensitive cells | 341.3 [202.1 to 430.2]
  Prednisolone-resistant cells | 447.9 [332.2 to 544.9]
Statistical Analysis 1: Comparison: Total Therapy; Test type: Superiority or Other; p = 0.00000095, Wilcoxon (Mann-Whitney)

7. Other Pre Specified Outcome: Median Difference in NLRP3 Gene Expression in Primary Leukemia Cells of Patients in Glucocorticoid-resistant Cells vs. Glucocorticoid-sensitive Cells
Description: Prednisolone sensitivity was measured in primary leukemia cells from bone marrow collected at diagnosis. Expression of NLRP3 was determined by HG-U133A microarray. Values given are gene expression values, and the unit is arbitrary units (AU) defined as scaled fluorescence measured on microarray.
Time Frame: Pre-treatment
Population: One hundred forty-four (144) patients were evaluable to assess prednisolone sensitivity measured in bone marrow ALL cells and NLRP3 expression in RNA by MTT assay
Measure: Median (Inter-Quartile Range); unit: arbitrary units
Arm/Group | Total Therapy
Number analyzed (Participants) | 144
arbitrary units
  Prednisolone-sensitive cells | 41.2 [31.4 to 58.7]
  Prednisolone-resistant cells | 110.7 [59.7 to 157.6]
Statistical Analysis 1: Comparison: Total Therapy; Test type: Superiority or Other; p = 0.0000007, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Participants were monitored from the start of therapy through 30 days after this protocol's treatment plan was completed.
Arm/Group | Total Therapy
Serious Adverse Events (participants affected / at risk) | 74/498
Other Adverse Events (participants affected / at risk) | 468/498
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Therapy (N=498)
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 2 (2)
Adult respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Allergic Reaction to Asparaginase (Immune system disorders) | 6 (6)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 2 (2)
Amylase (Metabolism and nutrition disorders) | 1 (1)
Apnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Bilirubin (Hepatobiliary disorders) | 1 (1)
CNS hemorrhage/bleeding (Blood and lymphatic system disorders) | 2 (2)
Catheter-related infection (Infections and infestations) | 3 (3)
Colitis (Gastrointestinal disorders) | 4 (4)
Creatinine (Renal and urinary disorders) | 1 (1)
DIC (disseminated intravascular coagulation) (Blood and lymphatic system disorders) | 2 (2)
Dermatology/Skin-Other (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema (General disorders) | 2 (2)
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (Infections and infestations) | 3 (4)
Fever (in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 10e9/L) (General disorders) | 3 (3)
Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Hepatic-Other (Hepatobiliary disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Cardiac disorders) | 2 (2)
Hypotension (Cardiac disorders) | 9 (9)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Infection (documented clinically or microbiologically) with grade 3 or 4 neutropenia (ANC <1.0 x 10e (Infections and infestations) | 32 (32)
Infection without neutropenia (Infections and infestations) | 5 (5)
Leukoencephalopathy associated with radiological findings (Nervous system disorders) | 2 (2)
Lipase (Metabolism and nutrition disorders) | 1 (1)
Liver dysfunction/failure (clinical), (Hepatobiliary disorders) | 2 (2)
Neuropathy-sensory (Nervous system disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 2 (2)
Personality/behavioral (Psychiatric disorders) | 1 (1)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary-Other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal failure (Gastrointestinal disorders) | 4 (4)
Seizure(s) (Nervous system disorders) | 6 (6)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Supraventricular arrhythmias (SVT/atrial fibrillation/flutter) (Cardiac disorders) | 1 (1)
Thrombosis/embolism (Cardiac disorders) | 5 (5)
Typhlitis (inflammation of cecum) (Gastrointestinal disorders) | 2 (2)
Vision-blurred vision (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Therapy (N=498)
Abdominal pain or cramping (General disorders) | 47 (69)
Allergic Reaction to Asparaginase (Immune system disorders) | 41 (45)
Anorexia (Gastrointestinal disorders) | 26 (31)
Catheter-related infection (Infections and infestations) | 86 (131)
Dehydration (Gastrointestinal disorders) | 29 (36)
Diarrhea patients without colostomy (Gastrointestinal disorders) | 53 (62)
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (Infections and infestations) | 436 (1407)
Fever (in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 10e9/L) (General disorders) | 208 (403)
Headache (General disorders) | 26 (38)
Hyperglycemia (Metabolism and nutrition disorders) | 43 (62)
Hypertension (Cardiac disorders) | 42 (42)
Hypokalemia (Metabolism and nutrition disorders) | 32 (36)
Hypotension (Cardiac disorders) | 52 (53)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 51 (62)
Infection (documented clinically or microbiologically) with grade 3 or 4 neutropenia (Infections and infestations) | 379 (893)
Infection without neutropenia (Infections and infestations) | 290 (594)
Neuropathic pain (Nervous system disorders) | 46 (46)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 35 (60)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 25 (25)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 29 (33)
SGPT (ALT) (Hepatobiliary disorders) | 76 (100)
Stomatitis/pharyngitis (oral/pharyngeal mucositis), (Gastrointestinal disorders) | 65 (75)
Thrombosis/embolism (Cardiac disorders) | 31 (34)
Typhlitis (Gastrointestinal disorders) | 27 (37)
Vomiting (Gastrointestinal disorders) | 59 (67)
Wound-infectious (Skin and subcutaneous tissue disorders) | 43 (48)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes